Protocol Title: Comparison of a Silicone Hydrogel Daily Disposable Multifocal Contact Lens to a Marketed Product

Protocol CR-6479

Version: 3.0

Date: 15 March 2022

Investigational Products: JJVC Investigational Multifocal Contact Lenses manufactured in senofilcon A C3

Keywords:

Senofilcon A C3, Delefilcon A, Presbyopia, Daily Wear, Daily Disposable, Dispensing, Randomized

#### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155:2020,<sup>1</sup> the International Council for Harmonization Good Clinical Practice E6(R2) (ICH GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

#### TABLE OF CONTENTS PROTOCOL TITLE, NUMBER, VERSION AND DATE......7 SPONSOR NAME AND ADDRESS.......7 AUTHORIZED SIGNATURES...... 8 CHANGE HISTORY 9 SYNOPSIS 10 COMMONLY USED ABBREVIATIONS. ACRONYMS AND DEFINITIONS OF TERMS 1.1. 1.2. 1.3. 1.4. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES ......21 2.1. 2.2. 2.3. 3.1. 3.2. 3.3. Exclusion Criteria 24 3.4. 4.1. Description of Study Design 26 4.2. 4.3. 5.1. 5.2. 5.3. 6.1. 6.2. Ancillary Supplies/Products 29

| 6.3. | Administration of Test Articles | 30 |
|-------|---------------------------------------------------|----|
| 6.4. | Packaging and Labeling | 30 |
| 6.5. | Storage Conditions | 30 |
| 6.6. | Collection and Storage of Samples | 30 |
| 6.7. | Accountability of Test Articles | 31 |
| 7. ST | TUDY EVALUATIONS | 32 |
| 7.1. | Time and Event Schedule | 32 |
| 7.2. | Detailed Study Procedures | 35 |
| Vl | ISIT 1 | 35 |
| Vl | ISIT 2 | 41 |
| Vl | ISIT 3 | 45 |
| Vl | ISIT 4 | 51 |
| Vl | ISIT 5 | 55 |
| Vl | ISIT 6 | 61 |
| FI | NAL EVALUATION | 63 |
| 7.3. | Unscheduled Visits | 64 |
| 7.4. | Laboratory Procedures | 65 |
| 8. SU | JBJECTS COMPLETION/WITHDRAWAL | |
| 8.1. | Completion Criteria | |
| 8.2. | Withdrawal/Discontinuation from the Study | 66 |
| 9. PF | RE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | |
| 9.1. | Systemic Medications | 67 |
| 10. | DEVIATIONS FROM THE PROTOCOL | 67 |
| | STUDY TERMINATION | |
| 12. 1 | PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 69 |
| 13. | ADVERSE EVENTS | 70 |
| 13.1. | Definitions and Classifications | 70 |
| 13.2. | Assessing Adverse Events | 72 |
| 13 | S.2.1. Causality Assessment | 72 |
| 13 | S.2.2. Severity Assessment | 73 |
| 13.3. | Documentation and Follow-Up of Adverse Events | 73 |
| 13.4. | Reporting Adverse Events | 75 |
| 13 | 4.1. Reporting Adverse Events to Sponsor | 75 |

| | 13.4.2 | <ol> <li>Reporting Adverse Events to the Responsible IEC/IRB and Health Author</li> <li>76</li> </ol> | orities |
|---|---|---|---|
| 13 | .5. | Event of Special Interest | 76 |
| 13 | .6. | Reporting of Pregnancy | 76 |
| 14. | STA | ATISTICAL METHODS | 76 |
| 14 | .1. | General Considerations | 76 |
| 14 | .2. | Sample Size Justification | 77 |
| 14 | .3. | Analysis Populations | 79 |
| 14 | .4. | Level of Statistical Significance | 79 |
| 14 | .5. | Primary Analysis | 79 |
| 14 | .6. | Secondary Analysis | 82 |
| 14 | .7. | Other Exploratory Analysis | 82 |
| 14 | .8. | Interim Analysis | 83 |
| 14 | .9. | Procedure for Handling Missing Data and Drop-Outs | 83 |
| 14 | .10. | Procedure for Reporting Deviations from Statistical Plan | 84 |
| 15. | DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | 84 |
| 15 | .1. | Electronic Case Report Form/Data Collection | 84 |
| 15 | .2. | Subject Record | 84 |
| 15 | .3. | Trial Registration on ClinicalTrials.gov | 85 |
| 16. | DA | TA MANAGEMENT | 85 |
| 16 | .1. | Access to Source Data/Document | 85 |
| 16 | .2. | Confidentiality of Information. | 85 |
| 16 | .3. | Data Quality Assurance | 85 |
| 16 | .4. | Data Monitoring Committee (DMC) | 86 |
| 17. | CL | NICAL MONITORING | 86 |
| 18. | ETI | HICAL AND REGULATORY ASPECTS | 86 |
| 18 | .1. | Study-Specific Design Considerations | 86 |
| 18 | .2. | Investigator Responsibility | 87 |
| 18 | .3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 87 |
| 18 | .4. | Informed Consent | 88 |
| 18 | .5. | Privacy of Personal Data | 88 |
| 19. | STU | JDY RECORD RETENTION | 89 |
| 20. | FIN | ANCIAL CONSIDERATIONS | 90 |
| 21. | PU | BLICATION | 90 |

| 22. REFERENCES | 91 |
|---|---|
| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 93 |
| APPENDIX B: PATIENT INSTRUCTION GUIDE | 100 |
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | 101 |
| APPENDIX D: PRESBYOPIC SYMPTOMS QUESTIONNAIRE | 104 |
| APPENDIX E: OCULAR DOMINANCE | 105 |
| APPENDIX F: LENS FITTING GUIDE | 106 |
| APPENDIX G: CONTROL LENS FITTING GUIDE | 108 |
| APPENDIX H: BINOCULAR OVER REFRACTION | 139 |
| APPENDIX I: | 140 |
| , Determination of Near Addition | 141 |
| , Near LogMAR Visual Acuity Measurement Procedure | 147 |
| , Lens Fitting Characteristics | 150 |
| , Subject Reported Ocular Symptoms/Problems | 156 |
| , Determination of Distance Spherocylindrical Refractive Error | 158 |
| , Biomicroscopy Scale | 164 |
| , Distance and Near Snellen Visual Acuity Evaluation | 170 |
| , Distance LogMAR Visual Acuity Measurement Procedure | 175 |
| , Patient Reported Outcomes | 179 |
| , Visual Acuity Chart Luminance and Room Illumination Testing | 181 |
| APPENDIX J: Guidelines for COVID-19 Risk Mitigation | 190 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 202 |
| LIST OF TABLES | |
| Table 1: Test Articles | |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | |
| Table 4: Disallowed systemic medications | |
| Table 5: Examples of major and minor protocol deviations | 68 |
| Table 6: Summary of Historical Studies Included in Sample Size Calculations | 77 |
| Table 7: Historical Odds Ratio Estimates and 95% CIs – Intent-to-Treat Population | |
| Table 8: Sample Size Estimates by Endpoint | |
| Table 9 Clinical Studies Planned to be Utilized in Exploratory Meta-Analysis | 83 |

| LIST OF FIGURES | |
|---------------------------|----|
| Figure 1: Study Flowchart | 16 |

#### PROTOCOL TITLE, NUMBER, VERSION AND DATE

Title: Protocol Title: Comparison of a Silicone Hydrogel Daily Disposable Multifocal Contact

Lens to a Marketed Product Protocol Number: CR-6479

Version: 3.0

Date: 15 March 2022

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care, Inc. (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR

| Name: |
|------------------------------|
| Title: |
| Address: |
| 24 Hour Contact Telephone #: |
| Email: |

The Medical Monitor must be notified by the clinical institution/site by e-mail or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

CR-6479, v 3.0

#### **AUTHORIZED SIGNATURES**

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, ISO 14155:2020, ICH guidelines, and the Declaration of Helsinki.

| Study Responsible<br>Clinician | |
|--------------------------------|---|
| Clinical Operations<br>Manager | |
| Biostatistician | |
| Data Management | |
| Reviewer | |
| Reviewer | |
| Medical Safety Officer | |
| Approver | _ |

#### **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and<br>Section Number(s) Affected | Justification for Change | Date |
|---|---|---|---|---|
| 1.0 | | Original Protocol | N/A | 30 Nov 2021 |
| 2.0 | | Throughout Document-<br>updated version number and<br>date. | Corrected<br>Typos | 03 Feb 2022 |
| | | Synopsis-corrected bullet numbering in inclusion. | | |
| | | Section 2.2-corrected bullet numbering. | | |
| | | Section 2.3-updated bullet numbering to match synopsis. | | |
| | | Section 7.1-T&E table removed wettability and deposits from table, removed PROs from V2 and V4 and added check for modifications at V3. | | |
| | | Section 14.7-added wording referring to Table 9. | | |
| 3.0 | | Throughout Document-<br>updated version number and<br>date. | Corrected<br>typo | 15 Mar 2022 |
| | | Section 7.2 step 1.9-corrected study lens to habitual lens. | | |

#### **SYNOPSIS**

| Protocol Title | Comparison of a Silicone Hydrogel Daily Disposable |
|---|---|
| Trotocor ritic | Multifocal Contact Lens to a Marketed Product |
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | |
| Cililical Filase | Clinical trial phase: Claims |
| Trial Desistantian | Design control phase: Phase 3 |
| Trial Registration | This study will be registered on ClinicalTrials.gov. |
| Test Article(s) | Investigational Product: JJVC Investigational Multifocal |
| | Contact Lenses manufactured in senofilcon A C3 (Aurora) |
| | Control: Dailies Total 1® Multifocal Contact Lenses |
| | manufactured in delefilcon A material (DT1MF) |
| Wear and Replacement | Wear Schedule: The test lenses will be used on a daily |
| Schedules | disposable basis. |
| | Replacement Schedule: The lenses will be replaced after a day |
| | of wear. |
| Objectives | Primary Objectives: |
| | The primary objective of this study is to compare the clinical |
| | performance of the JJVC Investigational Multifocal contact |
| | lens relative to Dailies Total-1 Multifocal (DT1MF) after 1- |
| | week of optimized lens wear with respect to subjective vision |
| | responses in low light vision and vision while reading in low |
| | light. |
| | Secondary Objectives: |
| | The secondary objective of this study is to compare the |
| | clinical performance of the JJVC Investigational Multifocal |
| | contact lens relative to Dailies Total-1 Multifocal (DT1MF) |
| | after 1-week of optimized lens wear with respect to distance, |
| | intermediate and near subjective vision responses. |

| | mison & Johnson Vision Care, Inc. |
|---|---|
| Study Endpoints | Co-primary endpoints: 1. Clarity of vision in dim or low lighting conditions [Item ID: P3_0006_p05] 2. Clarity of vision when reading in dim light (e.g., menu or bill in a restaurant [Item ID: P3_0006_p12]. |
| | <ol> <li>Secondary endpoints: <ol> <li>Clarity of distance vision (i.e., looking at things that are more than 5 feet away, such as street signs) [Item ID: P3_006_p10]</li> <li>Clarity of intermediate vision (i.e., looking at things 2-3 feet away, such as your computer screen) [Item ID: P3_006_p09]</li> <li>Clarity of near vision (i.e., looking at things close up, such as reading a book) [Item ID: P3_0006_p08]</li> </ol> </li> </ol> |
| | Other Endpoints: |
| | Group 1: Overall Opinion 1. Considering your experience with your current contact lenses, which statement best describes your overall opinion of these contact lenses? [Item ID: P3_0004_b00] |
| | <ul> <li>Group 2: Quality of Near Vision</li> <li>1. Blurred vision at close distances (such as reading a book) [Item ID: P3_0022_p01]</li> <li>2. Ease of re-focusing when you look from far to near [Item ID: P3_0006_p28]</li> <li>3. Clarity of vision when reading your cell phone [Item ID: P3_0006_p14]</li> </ul> |
| | <ul> <li>Group 3: Vision Consistency</li> <li>1. Consistent vision across all distance (near, far and inbetween) [Item ID: P3_0006_p26]</li> <li>2. Uninterrupted vision between and at all distances [Item ID: MIS01563]</li> <li>3. Clarity of vision during daily activities [Item ID: P3_0006_p04]</li> </ul> |
| | Group 4: 1. I experienced crisp clear vision at all distances [Item ID: MIS02043] 2. I experienced crisp clear vision in all lighting conditions [Item ID: MIS02044] |

conditions [Item ID: MIS02044]

| | Group 5: 1. Clarity of vision when reading your computer screen [Item ID: P3_0006_p15] |
|---|---|
| Study Design | This is a single-masked, 2×3 crossover, randomized-controlled, dispensing clinical trial. A total of approximately 110 eligible subjects will be targeted to complete the study. Subjects will be randomized and fit (Visit 1) in a study lens and wear the lens for 3±1 day then undergo optimization (Visit 2) and wear the optimized pair for approximately 1 week (7±1 day). At the follow-up visit (Visit 3) the endpoints will be measured and subjects will be fit in the 2 <sup>nd</sup> study lens. The visits will be repeated wearing the 2 <sup>nd</sup> study lens (Visit 3 Fit/Visit 4 Optimization/Visit 5 Follow up). At Visit 5 the subjects will be fit in a new pair of lenses that match the same type and power they were dispensed at Visit 4, and wear the lenses for 1 week (7±1 day). At the follow-up visit (Visit 6) the endpoints will be measured and the subject will be exited from the study. |
| | See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations. |
| Sample Size | A total of approximately 130 eligible subjects will be enrolled (78 myopes and 52 hyperopes) with 110 subjects (66 myopes and 44 hyperopes) targeted to complete. |
| Study Duration | The study will last approximately 2 to 3 months. |
| Anticipated Study | Healthy male and female volunteers with presbyopia will be |
| Population | screened as per criteria outlined below. All volunteers will |
| | have baseline measurements taken to ensure eligibility. The |
| | baseline procedures will occur after informed consent has |
| | been obtained. Subjects will have medical and contact lens |
| | history recorded, baseline questionnaires completed, and |
| | refractive and anterior segment status determined. For a detail flowchart of procedures below. |
| | Howehart of procedures below. |

# Eligibility Criteria - Potential subjects must satisfy all of the following criteria to be enrolled in the study

Inclusion Criteria after Screening:

The subject must:

- 1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Be at least 40 years of age and not greater than 70 years of age at the time of consent.
- 4. Own a wearable pair of spectacles if required for their distance vision.
- 5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month or more duration).
- 6. Either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" (Appendix D).

#### Inclusion Criteria at Baseline:

- 7. The subject's distance spherical equivalent refraction (vertex corrected if  $\geq$ -4.25 D) must be in the range of -1.25 D to -5.75 D or +0.75 D to +3.25 D in each eye.
- 8. The subject's refractive cylinder must be ≤0.75 D in each eye.
- 9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
- 10. The subject must have distance best corrected visual acuity of  $20/20^{-3}$  or better in each eye.

# Eligibility Criteria – Exclusion Potential subjects who meet any of the following criteria will be excluded from participating in the study: Exclusion Criteria after Screening: The subject must not:

- 1. Be currently pregnant or lactating.
- 2. Have any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
- 3. Have any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 4. Have any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, dacryocystorhinostomy, peripheral iridotomy/iridectomy, cataract surgery, retinal surgery, etc.).
- 5. Have a history of amblyopia, strabismus or binocular vision abnormality.
- 6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid, oral tetracyclines, anticholinergics, oral phenothiazines, oral/inhaled corticosteroids. See section 9.1 for further examples.
- 7. Use of any ocular medication, with the exception of rewetting drops.
- 8. Have a history of herpetic keratitis.
- 9. Have a history of irregular cornea.
- 10. Have a history of pathological dry eye.
- 11. Have Participated in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 12. Be and employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 13. Have any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.

Exclusion Criteria at Baseline: The subject must not:

| | <ul> <li>14. Have clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.</li> <li>15. Have any current ocular infection or inflammation.</li> <li>16. Have any current ocular abnormality that may interfere with contact lens wear.</li> </ul> |
|---|---|
| Disallowed<br>Medications/Interventions | Use of any prescription or over-the-counter (OTC) medications that may affect contact lens wear. See section 9.1 in the protocol for details regarding disallowed |
| | systemic medications. |
| Measurements and | logMAR acuity, subjective responses for vision, |
| Procedures | biomicroscopy and fit evaluations. |
| Microbiology or Other | None |
| Laboratory Testing | |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any serious adverse event (SAE) where relationship to study agent cannot be ruled out, may result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study- | |
| Specific Materials | ETDRS light cabinet, 4 M logMAR charts, and Near logMAR charts. |
| Principal Investigator(s) and Study Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



# COMMONLY USED ABBREVIATIONS, ACRONYMS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager
COVID-19 Coronavirus Disease 2019
CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDEInvestigational Device ExemptionIECIndependent Ethics CommitteeIRBInstitutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NAVQ Near Activity Visual Questionnaire

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye
OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

The purpose of this study is to evaluate the subjective responses of the JJVC Investigational Multifocal Contact Lens. The Test lenses are silicone hydrogel daily disposable contact lenses. The performance of these new lenses will be compared to a marketed product, Dailies Total 1<sup>®</sup> Multifocal Contact Lenses.

#### 1.1. Name and Descriptions of Investigational Products

Investigational Product: JJVC Investigational Multifocal Contact Lenses manufactured in senofilcon A C3

Control: Dailies Total 1<sup>®</sup> Multifocal Contact Lenses manufactured in delefilcon A material

#### 1.2. Intended Use of Investigational Products

All lenses are intended to correct spherical refractive error and presbyopia. For this study both of the lenses will be worn as a daily disposable lens, with the lenses being discarded after a day of wear. The Lenses will be fit in a randomized fashion. After fitting, each subject will return for an optimization visit and then a follow-up.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding the Test lenses refer to the latest version of the CR-6479 Investigational Brochure.<sup>5</sup>

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

Anticipated risks and adverse reactions with this lens are similar to those with other soft daily wear contact lenses used to correct presbyopia. A listing of examples of adverse reactions is found in the section 13 of this protocol. The investigator should follow normal clinical guidelines regarding examination and care of subjects who participate in this trial. Refer to study lens package insert for additional details for the control lens and the Investigational Brochure (IB) for the Investigational lens.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study



CR-6479, v 3.0



was a single masked, randomized controlled, dispensing clinical trial on myopic presbyopes and had a primary endpoint of logMAR visual acuity. There were 66 subjects that completed the study per the protocol. The lenses displayed good clinical vision performance with binocular, high luminance, high contrast logMAR visual acuity of -0.128, -0.061 and 0.057 at distance, intermediate and near respectively. There was one adverse of event during the study. The one ocular adverse event was a non-significant grade 2 or less slit lamp finding requiring treatment. The event was classified as related and occurred while wearing the control lens.<sup>13</sup>

For information about the control product refer to study lens package insert for additional details (APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) and the Investigational Brochure (IB) for the Investigational product.<sup>5</sup>

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

#### Primary Objective:

The primary objective of this study is to compare the clinical performance of the JJVC Investigational Multifocal contact lens (Test) relative to Dailies Total-1 Multifocal contact lens (DT1MF) after 1-week of optimized lens wear with respect to subjective vision responses in low light vision and vision while reading in low light.

#### Secondary Objective:

The secondary objective of this study is to compare the clinical performance of the Test lens relative to the DT1MF lens after 1-week of optimized lens wear with respect to subjective vision responses related to clarity of distance, intermediate and near vision.

#### 2.2. Endpoints

#### Co-Primary Endpoints:

- 1. Clarity of vision in dim or low lighting conditions [Item ID: P3 0006 p05]
- 2. Clarity of vision when reading in dim light (e.g., menu or bill in a restaurant [Item ID: P3 0006 p12].

#### Secondary Endpoints:

- 1. Clarity of distance vision (i.e., looking at things that are more than 5 feet away, such as street signs) [Item ID: P3\_006\_p10]
- 2. Clarity of intermediate vision (i.e., looking at things 2-3 feet away, such as your computer screen) [Item ID: P3 006 p09]
- 3. Clarity of near vision (i.e., looking at things close up, such as reading a book) [Item ID: P3\_0006\_p08]

Co-primary and secondary endpoints will be assessed at the 1-week follow-up evaluation (in the optimized lenses) using individual questionnaire items. Co-primary and secondary endpoints will utilize an Excellence response set (0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor).

#### **Exploratory Endpoints:**

#### Group 1: Overall Opinion

1. Considering your experience with your current contact lenses, which statement best describes your <u>overall opinion</u> of these contact lenses? [Item ID: P3\_0004\_b00]

#### Group 2: Quality of Near Vision

- 1. Blurred vision at close distances (such as reading a book) [Item ID: P3\_0022\_p01]
- 2. Ease of re-focusing when you look from far to near [Item ID: P3 0006 p28]
- 3. Clarity of vision when reading your cell phone [Item ID: P3 0006 p14]

#### Group 3: Vision Consistency

- 1. Consistent vision across all distance (near, far and in-between) [Item ID: P3 0006 p26]
- 2. Uninterrupted vision between and at all distances [Item ID: MIS01563]
- 3. Clarity of vision during daily activities [Item ID: P3\_0006\_p04]

#### Group 4:

- 1. I experienced crisp clear vision at all distances [Item ID: MIS02043]
- 2. I experienced crisp clear vision in all lighting conditions [Item ID: MIS02044]

#### Group 5:

1. Clarity of vision when reading your computer screen [Item ID: P3 0006 p15]

All exploratory endpoints will be assessed at the 1-week follow-up evaluation (in the optimized lenses) using individual questionnaire items. Exploratory group 1 overall opinion will utilize the following Excellence response set (1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor). For both group 2 (endpoints 2 and 3) and group 3 (all endpoints) the following Excellence response set will be used (0: Not Applicable, 1: Excellent, 2: Very Good, 3: Good, 4: Fair and 5: Poor). With respect to endpoint 1 within group 2, the following Frequency response set will be used (1: Always, 2: Frequently, 3: Occasionally, 4: Rarely, 5: Never and 6: Don't Know). Group 4 will utilize the following Agreement response set (1: Agree Strongly, 2: Agree Somewhat, 3: Neither Agree Nor Disagree, 4: Disagree Somewhat and 5: Disagree Strongly).

#### 2.3. Hypotheses

All primary and secondary hypotheses must be met in order to satisfy the objective of this study.

#### Co-Primary Hypotheses

- 1. After approximately 1-week of wear in the optimized lenses, the Test lens will be superior to DT1MF with respect to clarity of vision in dim or low lighting conditions.
- 2. After approximately 1-week of wear in the optimized lenses, the Test lens will be superior to DT1MF with respect to clarity of vision when reading in dim light.

Both co-primary hypotheses must be met prior to testing the secondary hypotheses.

#### Secondary Hypotheses

- 1. After approximately 1-week of wear, the Test lens will be non-inferior to DT1MF with respect to clarity of distance vision. A non-inferiority margin of 10% will be used.
- 2. After approximately 1-week of wear, the Test lens will be superior to DT1MF with respect to clarity of intermediate vision.
- 3. After approximately 1-week of wear, the Test lens will be superior to DT1MF with respect to clarity of near vision.

All primary and secondary hypotheses must be met in order to test any exploratory hypotheses.

#### **Exploratory Hypotheses**

1. After 1-week of wear in the optimized lenses, the Test lens will be superior to DT1MF with respect to each of the following:

#### Group 1:

1. Overall Opinion

#### Group 2:

- 1. Blurred vision at close distances
- 2. Ease of re-focusing when you look from far to near
- 3. Clarity of vision when reading your cell phone

#### Group 3:

- 1. Consistent vision across all distance
- 2. Uninterrupted vision between and at all distances
- 3. Clarity of vision during daily activities

#### Group 4:

- 1. I experienced crisp clear vision at all distances
- 2. I experienced crisp clear vision in all lighting conditions

#### Group 5:

1. Clarity of vision when reading your computer screen

If exploratory hypotheses are tested, historical data will be combined with the current study data for the statistical analysis. See section 14 for more information.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Healthy male and female subjects who are habitual soft contact lens wearers will be recruited. Subjects will be at least 40 years of age and not older than 70 years of age. Subjects enrolled in this study will be either myopic or hyperopic and have presbyopia.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all the following criteria to be enrolled in the study:

Inclusion Criteria after Screening:

The subject must:

- 1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Be at least 40 years of age and not greater than 70 years of age at the time of consent.
- 4. Own a wearable pair of spectacles if required for their distance vision.
- 5. Be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 6 hours per wear day, for 1 month or more duration).
- 6. Either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" (Appendix D).

#### Inclusion Criteria at Baseline:

- 7. The subject's distance spherical equivalent refraction (vertex corrected if  $\geq$ -4.25 D) must be in the range of -1.25 D to -5.75 D or +0.75 D to +3.25 D in each eye.
- 8. The subject's refractive cylinder must be  $\leq 0.75$  D in each eye.
- 9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
- 10. The subject must have distance best corrected visual acuity of 20/20<sup>-3</sup> or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria after Screening:

The subject must not:

- 1. Be currently pregnant or lactating.
- 2. Have any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
- 3. Have any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 4. Have any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, dacryocystorhinostomy, peripheral iridotomy/iridectomy, cataract surgery, retinal surgery, etc.).
- 5. Have a history of amblyopia, strabismus or binocular vision abnormality.
- 6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid, oral tetracyclines, anticholinergics, oral phenothiazines, oral/inhaled corticosteroids. See section 9.1 for further examples.
- 7. Use of any ocular medication, with the exception of rewetting drops.
- 8. Have a history of herpetic keratitis.
- 9. Have a history of irregular cornea.
- 10. Have a history of pathological dry eye.
- 11. Have Participated in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 12. Be and employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 13. Have any known hypersensitivity or allergic reaction to non-preserved rewetting drop solutions or sodium fluorescein.

Exclusion Criteria at Baseline:

The subject must not:

- 14. Have clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 15. Have any current ocular infection or inflammation.
- 16. Have any current ocular abnormality that may interfere with contact lens wear.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

This is a 6-visit, single-masked, multi-site 2×3 crossover, randomized-controlled, dispensing clinical trial. A total of approximately 130 eligible subjects will be enrolled (78 myopes and 52 hyperopes) with 110 subjects (66 myopes and 44 hyperopes) targeted to complete.

At the initial visit (Visit 1), if a subject is found to meet all eligibility criteria, they will be randomized to one of two lens wear sequences and fitted with the first study lens; otherwise, the subject will be deemed ineligible and classified as a screen failure.

Subjects will be dispensed their first lens per the randomization schedule at Visit 1 and wear the lens for 3±1 day. Subjects will return for Visit 2 and then undergo optimization and wear the optimized lens pair for approximately 1 week (7±1 day). At the follow-up visit (Visit 3), endpoints will be measured and subjects will be fit in their 2nd study lens per the randomization scheme. Subjects will return approximately 3±1 day for Visit 4 and undergo lens optimization for the end lens. The optimized lens pair for the 2<sup>nd</sup> study lens will be worn for approximately 1 week (7±1 day). Subjects will return for Visit 5, the same study endpoints as Visit 3 will be measured and subjects will be fit and dispensed their 3<sup>rd</sup> study lens. Subjects will wear the 3<sup>rd</sup> study lens for 1 week (7±1 day) and return for the follow-up visit (Visit 6) the endpoints will be measured and the subject will be exited from the study.

Subjects will be advised to wear the study lenses every day while they are in the study for a minimum of 6 hours per day. The study lens will be replaced at the optimization visit. However, lost or damaged lenses may be replaced when necessary. Unscheduled visit may be conducted.

#### 4.2. Study Design Rationale

Crossover designs are a well-established study design in which subjects are exposed to multiple treatments during different time periods. A 2×3 bilateral crossover design was considered to be the optimal design since the study period is relatively short, the design can be cost effective, and more efficient comparisons between treatments can be made. As compared to a parallel study since fewer subjects are required to achieve the same pre-specified statistical power. Each subject will act as their own control to reduce the influence of potential confounding factors such as age, gender and vision correction.

#### 4.3. Enrollment Target and Study Duration

A total of approximately 130 eligible subjects will be enrolled (78 myopes and 52 hyperopes) will be enrolled with 110 subjects (66 myopes and 44 hyperopes) targeted to complete. The study is anticipated to last 2-3 months.


#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn in a bilateral and random fashion using a 2x3 crossover design. A computer-generated randomization scheme will be used to randomly assign subjects, in blocks of 2, to one of the two lens wear sequences: Test/DT1MF/DT1MF or DT1MF/Test/Test. The randomization scheme will be stratified by site. The random scheme will be generated using the PROC PLAN procedure from Statistical Analysis System (SAS) Software Version 9.4 or higher (SAS Institute, Cary, NC).<sup>15</sup>

The study site must follow the randomization scheme provided and complete enrollment per the randomization list and not pre-select or assign subjects. Randomization will be performed at visit first visit prior to the first fitting. The following must have occurred prior to randomization:

- Informed consent must have been obtained.
- The subject must have met all eligibility criteria.
- The subject's screening and baseline information must have been collected.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule to obtain the test article assignment for that subject prior to dispensing.
- 2. Investigator or designee will record the subject's number on the appropriate line of the lens fitting schedule.
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section.

#### 5.2. Masking

This is a single-masked study. Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

#### 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing.
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme if applicable

Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| Table 1. Test Afficies | Toot | Control |
|---|---|---|
| 37 | Test | Control |
| Name | JJVC Investigational | Dailies Total 1® Multifocal |
| | Multifocal Contact Lens | Contact Lens |
| Manufacturer | Johnson & Johnson® Vision | Alcon |
| | Care, Inc. | |
| | | N/A |
| Lens Material | senofilcon A (C3) | delefilcon A |
| Nominal Base Curve | 8.35 mm/8.5 mm (sphere) | 8.5 mm |
| Nominal Diameter | 14.3 mm | 14.1 mm |
| Nominal Distance | -1.00 D to | -0.75 D to -6.00 D and +0.50 D |
| Powers (D) | -6.00 D and +0.50 D to | to +3.75 D in 0.25 D steps |
| | +3.50 D in 0.25 D steps | |
| Nominal ADD Powers | LOW, MID, HI | LO, MED, HI |
| (D) | | |
| W | 200/ | 220/ |
| Water Content | 38% | 33% |
| Center Thickness | Varies with power | Varies with power |
| Oxygen Permeability | 103 | 156 |
| (Dk) | | |
| Wear Schedule in | Daily Wear | Daily Wear |
| Current Study | | |
| Replacement Frequency | Daily | Daily |
| Packaging Form (vial, | Blister | Blister |
| blister, etc.) | | |
| Packaging Form (vial, | Blister | Blister |
| blister, etc.) | | |

#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Single-Use Preservative-Free Rewetting Solutions (any one | | |
|---|---|---|---|
| | of these three rewetting solutions options may be supplied) | | |
| | Eye-Cept <sup>®</sup> | ScleralFil <sup>®</sup> | LacriPure Saline |
| Solution Name/Description | Rewetting Drops | Preservative Free | Solution |
| _ | | Saline Solution | |
| Manufacturer | Optics Laboratory | B&L | Menicon |
| Preservative | Non-Preserved | Non-preserved | Non-preserved |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the investigator and/or the sponsor.

#### 6.4. Packaging and Labeling

The test articles will be packaged in blisters, as the primary packaging. The test article will be over-labeled to mask the subject to the identity of the lens. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:



#### **6.5.** Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Event and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

CR-6479, v 3.0

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- 2. What was returned to the Investigator unused, including expired or malfunctioning product.
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

Reference : Site Instructions for Test Article Receipt and Test Article Accountability for additional information.

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1<br>Screening,<br>Baseline,<br>Treatment | Visit 2<br>Treatment 1<br>Follow-up 1<br>Optimization | Visit 3 Treatment 1 Follow-up 2, Treatment 2 | Visit 4 Treatment 2 Follow-up 1, Optimizati on | Visit 5 Treatment 2 Follow-up 2, Treatment 3 | Visit 6 Treatment 3 Follow-up 1 |
|---|---|---|---|---|---|---|
| Time Point | Day 0 | Day 3±1<br>from V1 | Day 7±1<br>from V2<br>Day 0 | Day 3±1<br>from V3 | Day 7±1<br>from V4 | Day 7±1<br>from V5 |
| Estimated Visit<br>Duration | 2.5 hours | 1.0 hour | 2.0 hour | 1.0 hour | 2.0 hour | 1.5 hour |
| Statement of | | | | | | |
| Informed Consent | X | | | | | |
| Demographics | X | | | | | |
| Medical | | | | | | |
| History/Concomitant | x | | | | | |
| Medications | | | | | | |
| Adverse Events and | | | | | | |
| Concomitant | | X | X | X | X | X |
| Medications Review | | | | | | |
| Compliance | | X | X | X | X | X |
| Habitual Contact | | | | | | |
| Lens Information | X | | | | | |
| Contact Lens History | х | | | | | |
| Wear Time and | | | | | | |
| Comfortable Wear | | | | | | |
| Time with Habitual | X | | | | | |
| lenses | | | | | | |
| Wear Time and | | | | | | |
| Comfortable Wear | | | T- | | | |
| Time with Study | | X | X | X | X | X |
| lenses | | | | | | |
| Screening | | | | | | |
| Inclusion/Exclusion | X | | | | | |
| Criteria | | | | | | |
| Subject Reported | | | | | | |
| Ocular Symptoms | X | X | X | X | X | X |
| Baseline PRO | | | | | | |
| (MRD) | X | | | | | |
| Questionnaire | | | | | | |

| Visit Information | Visit 1<br>Screening,<br>Baseline,<br>Treatment | Visit 2<br>Treatment 1<br>Follow-up 1<br>Optimization | Visit 3 Treatment 1 Follow-up 2, Treatment 2 | Visit 4 Treatment 2 Follow-up 1, Optimizati on | Visit 5 Treatment 2 Follow-up 2, Treatment 3 | Visit 6 Treatment 3 Follow-up 1 |
|---|---|---|---|---|---|---|
| Time Point | Day 0 | Day 3±1<br>from V1 | Day 7±1<br>from V2<br>Day 0 | Day 3±1<br>from V3 | Day 7±1<br>from V4 | Day 7±1<br>from V5 |
| Estimated Visit Duration | 2.5 hours | 1.0 hour | 2.0 hour | 1.0 hour | 2.0 hour | 1.5 hour |
| Distance and Near<br>Entrance Visual<br>Acuity | X | X | X | х | X | х |
| Lens Removal | X | X | X | X | X | X |
| Subjective Refraction and Distance Visual Acuity | Х | | | | | |
| Near ADD Determination | X | | | | | |
| Ocular Dominance | X | | | | | |
| ADD Refinement | X | | | | | |
| Near Visual Acuity | X | | | | | |
| Biomicroscopy | X | X | X | X | X | X |
| Baseline Inclusion/<br>Exclusion Criteria | X | | | | | |
| Continuance | | | X | | X | |
| Lens Selection | X | x (if<br>modified) | X | x (if<br>modified) | X | |
| Lens Insertion | X | X | X | X | X | |
| 10-Minute Settling | X | x (if<br>modified) | | x (if modified) | X | |
| Visual Satisfaction / Subjective Acceptance | X | Х | X | X | X | х |
| Study Lens Distance<br>and Near Visual<br>Acuity | X | х | Х | Х | X | х |
| Distance Over<br>Refraction and<br>Visual Acuity | X | х | Х | X | X | х |
| Subjective Lens Fit<br>Assessment | X | х | X | X | X | X |
| Binocular Over<br>Refraction | | | X | | X | Х |

| Visit Information | Visit 1<br>Screening,<br>Baseline,<br>Treatment | Visit 2<br>Treatment 1<br>Follow-up 1<br>Optimization | Visit 3 Treatment 1 Follow-up 2, Treatment 2 | Visit 4 Treatment 2 Follow-up 1, Optimizati on | Visit 5 Treatment 2 Follow-up 2, Treatment 3 | Visit 6 Treatment 3 Follow-up 1 |
|---|---|---|---|---|---|---|
| Time Point | Day 0 | Day 3±1<br>from V1 | Day 7±1<br>from V2<br>Day 0 | Day 3±1<br>from V3 | Day 7±1<br>from V4 | Day 7±1<br>from V5 |
| Estimated Visit<br>Duration | 2.5 hours | 1.0 hour | 2.0 hour | 1.0 hour | 2.0 hour | 1.5 hour |
| Compliance | | Х | X | Х | Х | х |
| Follow-up PRO<br>(MRD)<br>Questionnaire | | | x | | x | х |
| Visual Performance | | | X | | Х | X |
| Modifications | X | X | X | X | | |
| Distance and Near<br>Exit Visual Acuity | X | х | X | X | X | |
| Dispensing Criteria | X | X | X | X | X | |
| Instructions | X | X | X | X | X | |
| Schedule Follow-up | X | X | X | X | X | |
| Final Evaluation | | | | | | X |

#### 7.2. Detailed Study Procedures

#### VISIT 1

Subjects must report to the visit wearing their habitual contact lenses to accurately assess baseline PRO (MRD) performance. If the subject is not wearing their lenses they must be rescheduled.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. NOTE: The subject must be provided a signed copy of this document. |
| 1.2 | Demographics | Record the subject's age, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subject's medical history and concomitant medications. |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |
| 1.5 | Habitual Lens Duration of Wear/Days per week | Questions regarding the subject's duration of contact lens wear and the minimum number of days they wear their lenses per week. |
| 1.6 | Contact Lens History | Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). |
| 1.7 | Wear time and<br>Comfortable Wear<br>time with Habitual<br>lenses | Record the subject's wear time and comfortable wear time with their habitual contact lenses. |
| 1.8 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms are not required. |

| | Visit 1: Baseline | | | | | |
|---|---|---|---|--|--|--|
| Step | Procedure | Details | | | | |
| 1.9 | Baseline PRO<br>(MRD)<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, and visual symptoms of their habitual lenses using the PRO (MRD) questionnaires. | | | | |
| 1.10 | Ocular Symptoms | The subject will respond to a verbal openended symptoms questionnaire. | | | | |
| 1.11 | Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the subject's habitual contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | | | | |
| 1.12 | Lens Removal | Have the subject remove their habitual lenses and store in an approved storage solution. | | | | |
| 1.13 | Subjective<br>Refraction and<br>Distance Visual<br>Acuity | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity to the nearest letter. NOTE: Best distance visual acuity with sphero-cylindrical refraction must be at least 20/20 <sup>-3</sup> in each eye for the subject to be eligible in the study. | | | | |
| 1.14 | Near ADD Determination | The near reading addition will be determined using the binocular crossed cylinder technique (BCC) at 40 cm. | | | | |
| 1.15 | Ocular Dominance | Determine the distance ocular dominance with the best distance correction in place using a +1.00-blur test. If the results are equivocal use the sighting dominance test to determine the dominant eye used for the study. | Appendix<br>E | | | |
| 1.16 | ADD Refinement | Place the BCC result in the trial frame and refine the near prescription with trial lenses (or flippers) under binocular conditions. | | | | |
| 1.17 | Near Visual Acuity | Using the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm. Record the near visual acuity OD, OS and OU at 40 cm. | | | | |
| | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.18 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. | |
| | | If any of these slit lamp findings are Grade 2 or higher, the subject will be discontinued. If discontinued a final examination must be completed. | |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. | |
| 1.19 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. If so, proceed to lens fitting. | |
| | | If subject is deemed to be ineligible after baseline, proceed to Final Evaluation and complete all forms. | |
| | | Visit 1: Treatment 1 Lens Fitting | |
| Step | Procedure | Details | |
| 1.20 | Randomization | Record the randomization ID. | |
| 1.21 | Lens Selection | Select the lens pair and power based on the randomization scheme, spherical equivalent refraction and fitting guide for each eye. Record the Test lens parameters (power and lot number). | Appendix F or G (Fitting Guide) |
| 1.22 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated from the other worn lenses that will be | |
| 1.00 | | shipped back to the Sponsor. Complete the Product Quality Complaint form. | |
| 1.23 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. | |
| 1.24 | Determine Visual Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject | |

| | Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | to look down a hallway or out of a window<br>for distance vision assessments, and for them<br>to read a book, magazine or similar for near<br>vision. | |
| 1.25 | Study Lens Distance<br>and Near Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. Note: Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity | |
| 1.26 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 1.27 | Modifications | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted, if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 1.22-1.27 will be repeated for each modification. | Appendix F or G (Fitting Guide) |
| 1.28 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). | |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | The subject should not proceed to wear the lenses if any of the following is observed: |
| | | <ul> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze and push-up)</li> </ul> |
| | | NOTE: If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses and complete the Final Evaluation forms. |
| 1.29 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| | | <u>NOTE</u> : The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. |
| 1.30 | Dispensing Criteria | <ul> <li>The following criteria must be met for lenses to be dispensed and if all are not met the subject will be discontinued.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is</li> </ul> |
| | | <ul> <li>acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |
| 1.31 | Patient Instructions | <ul><li>Instruct the Subject the following:</li><li>The lenses will be worn on a daily wear basis.</li></ul> |

| | | Visit 1: Treatment 1 Lens Fitting |
|---|---|---|
| Step | Procedure | Details |
| Step | Procedure | <ul> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> <li>NOTE: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the</li> </ul> |
| 1.32 | Schedule | Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. The subject will be scheduled to return for |
| | Follow-up | their follow-up appointment in 3±1 days. |

| | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | NOTE: To count the follow-up visit as a day |
| | | of wear the Subject must have worn the |
| | | study lenses for 6 hours prior to the visit. |

#### VISIT 2

The subjects must present to Visit 2 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 2: Treatment 1 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 2.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 2.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 2.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for at least 6 hours per day. To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 2.4 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 2.5 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 2.6 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity |
| 2.7 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record |

| | Visit 2: Treatment 1 Follow-up 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | the results and distance visual acuity OD and OS. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 2.8 | Determination of Lens Optimization | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide and steps 1.22-1.27 in Visit 1 Fitting allowing for at least 10 minutes of settling time between each lens modification. | Appendix F or G (Fitting Guide) |
| 2.9 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). | |

| | Visit 2: Treatment 1 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | <u>NOTE</u> : If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses and complete the Final Evaluation forms. |
| 2.10 | Collection of<br>unworn lenses (if<br>applicable) | Collect unworn lenses returned by the subject when lens power has been optimized. If lens power was not changed allow the subject to use the unworn lenses dispensed at Visit 1 and dispense enough lenses of the same power to last the subject until their next visit. |
| 2.11 | Lens Removal | The study lenses will be removed and discarded. |
| 2.12 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative free rewetting drops |
| | | expedited, preservative-free rewetting drops may be instilled. |
| 2.13 | Insertion of Study<br>Lenses | Dispense the subject a new pair of lenses that match the distance and ADD power of the lenses that were removed in Step 2.11 above. |
| 2.14 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. NOTE: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. |
| 2.15 | Dispensing Criteria | <ul> <li>The following criteria must be met for lenses to be dispensed and if all are not met the subject will be discontinued.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> </ul> |

| | Visit 2: Treatment 1 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | Lenses must have an acceptable general lens fit. |
| 2.16 | Patient Instructions | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>NOTE: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor.</li> </ul> |

| | Visit 2: Treatment 1 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 2.17 | Schedule | The subject will be scheduled to return for |
| | Follow-up | their follow-up appointment in 7±1 days. |
| | | <u>NOTE</u> : To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

#### VISIT 3

The subjects must present to Visit 3 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 3: Treatment 1 Follow-up 2 | |
|---|---|---|
| Step | Procedure | Details |
| 3.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 3.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 3.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for at least 6 hours per day. To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 3.4 | PRO (MRD)<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, and visual symptoms of the study lenses using the PRO (MRD) questionnaires. |
| 3.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire |
| 3.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 3.7 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be |

| | Visit 3: Treatment 1 Follow-up 2 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | recorded to the nearest letter OD, OS and OU. | |
| 3.8 | Visual Performance<br>Distance (4M)<br>Intermediate (64 cm)<br>Near (40 cm) | Binocular Visual performance will be recorded for the following: Distance, Bright Illuminance High and Low Contrast ETDRS Charts 4M-HC#3 and LC#3 | |
| | | Near, Bright Illuminance Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast and Low Contrast Near (40 cm) High Contrast and Low Contrast | |
| | | <ul> <li>Note:</li> <li>The room illuminance must be between 7.3 and 7.9 EV (394-597 lux).</li> <li>Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV (181-208 cd/m²).</li> <li>Guillon-Poling, Near Chart Luminance Acceptable Range 10.8-11.1 EV (223-274 cd/m²).</li> </ul> | |
| 3.9 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix H |
| 3.10 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift | |

| | Visit 3: Treatment 1 Follow-up 2 | |
|---|---|---|
| Step | Procedure | Details |
| | | presence of unacceptable movement<br>(excessive or insufficient) in <u>all three</u><br>movement categories (primary gaze,<br>upgaze, and push-up). |
| | | <u>NOTE</u> : If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses and complete the Final Evaluation forms. |
| 3.11 | Collection of unworn lenses (if applicable) | Collect unworn lenses returned by the subject. |
| 3.12 | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. NOTE: Lenses do not need to be stored in a refrigerator. |
| 3.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 3.14 | Continuance | Determine whether the subject is eligible to continue in the study based on the examination findings. |

| | Visit 3: Treatment 2 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 3.15 | Lens Selection | Select the lens pair and power based on the randomization scheme, spherical equivalent refraction (measured at Visit 1 baseline) and fitting guide for each eye. Record the Test lens parameters (power and lot number). | Appendix F or G (Fitting Guide) |
| 3.16 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated from the other worn lenses that will be | |

| | | Visit 3: Treatment 2 Lens Fitting | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | shipped back to the Sponsor. Complete the | |
| | | Product Quality Complaint form. | |
| 3.17 | Lens Settling | Allow the study lenses to settle for a | |
| | | minimum of 10 minutes. | |
| 3.18 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. | |
| 3.19 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 3.20 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 3.21 | Modifications | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted, if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. | Appendix F or G (Fitting Guide) |

| | 7 | Visit 3: Treatment 2 Lens Fitting |
|---|---|---|
| Step | Procedure | Details |
| | | If modifications are required steps 3.20-3.25 will be repeated for each modification. |
| 3.22 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). |
| | | The subject should not proceed to wear the lenses if any of the following is observed: |
| | | <ul> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> </ul> |
| | | presence of unacceptable movement<br>(excessive or insufficient) in <u>all three</u><br>movement categories (primary gaze,<br>upgaze, and push-up). |
| | | NOTE: If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses and complete the Final Evaluation forms. |
| 3.23 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| | | <u>NOTE</u> : The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. |
| 3.24 | Dispensing Criteria | The following criteria must be met for lenses to be dispensed and if all are not met the subject will be discontinued. |
| | | <ul> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is</li> </ul> |
| | | acceptable. |
| | | • Subject must indicate that the comfort of the lenses is acceptable. |

| | Visit 3: Treatment 2 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | Lenses must have an acceptable general lens fit. |
| 3.25 | Patient Instructions | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> </ul> |
| | | NOTE: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn |

| | Visit 3: Treatment 2 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | lenses that will be shipped back to the |
| | | Sponsor. |
| 3.26 | Schedule | The subject will be scheduled to return for |
| | Follow-up | their follow-up appointment in 3±1 days. |
| | | <u>NOTE</u> : To count the follow-up visit as a day |
| | | of wear the Subject must have worn the |
| | | study lenses for 6 hours prior to the visit. |

#### VISIT 4

The subjects must present to Visit 4 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 4: Treatment 2 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 4.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 4.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses Wear Time | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 4.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 4.4 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 4.5 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 4.6 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. |

| | Visit 4: Treatment 2 Follow-up 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| | | Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity | |
| 4.7 | Distance Over-Refraction and Distance Visual Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results and distance visual acuity OD and OS. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 4.8 | Determination of Lens Optimization | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted, if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide and steps 3.20-3.25 in Visit 3 Fitting allowing for at least 10 minutes of settling time between each lens modification. | Appendix F<br>or G<br>(Fitting<br>Guide) |
| 4.9 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift | |

| | Visit 4: Treatment 2 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | presence of unacceptable movement (excessive or insufficient) in <u>all three</u> movement categories (primary gaze, upgaze, and push-up). <u>NOTE</u> : If lens fit is unacceptable subject |
| | | will be discontinued from the study. Remove the lenses and complete the Final |
| | | Evaluation forms. |
| 4.10 | Collection of unworn lenses (if applicable) | Collect unworn lenses returned by the subject when lens power has been optimized. If lens power was not changed allow the |
| | | subject to use the unworn lenses dispensed at Visit 3 and dispense enough lenses of the same power to last the subject until their next visit. |
| 4.11 | Lens Removal | The study lenses will be removed and discarded. |
| 4.12 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit<br>Lamp Classification Scales will be used to<br>grade the findings. |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 4.13 | Insertion of Study<br>Lenses | Dispense the subject a new pair of lenses that match the distance and ADD power of the lenses that were removed in Step 4.11 above. |
| 4.14 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| | | <u>NOTE:</u> The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. |
| 4.15 | Dispensing Criteria | The following criteria must be met for lenses to be dispensed and if all are not met the subject will be discontinued. |

| | Visit 4: Treatment 2 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | <ul> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> </ul> |
| | | <ul> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |
| 4.16 | Patient Instructions | Instruct the Subject the following: The lenses will be worn on a daily wear basis. Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed. A new lens will be opened and worn each day. Instruct the subject to bring back all unworn study lenses. Instruct the subject no cleaning or disinfecting solutions will be used for this lens type. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness. Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study. Subjects will be instructed to wear their glasses when not wearing the study lenses. NOTE: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if |

| | Visit 4: Treatment 2 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| | | possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. |
| 4.17 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 days. NOTE: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

#### VISIT 5

The subjects must present to Visit 5 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| Visit 5: Treatment 2 Follow-up 2 | | |
|---|---|---|
| Step | Procedure | Details |
| 5.1 | Adverse Events and | Review the subject's concomitant |
| | Concomitant | medications and record any changes from the |
| | Medications Review | previous study visit. |
| | | Record any adverse events or medical history |
| | | changes from the previous study visit. |
| 5.2 | Wear time and | Record the hours the subject has worn the |
| | Comfortable Wear | study lenses and the comfortable wear time |
| | time with Study | on the day of follow-up. |
| | lenses | |
| 5.3 | Compliance | Record the subject's compliance with |
| | | wearing the study lenses. |
| | | NOTE: Subjects must be made long as for |
| | | <u>NOTE</u> : Subjects must have worn lenses for at least 6 hours per day |
| | | To be counted as a day of wear at this visit |
| | | the Subject must have worn the study lenses |
| | | for 6 hours prior to the visit. |
| 5.4 | PRO (MRD) | The subject will evaluate the vision |
| 3.4 | Questionnaires | characteristics, comfort characteristics, and |
| | Questionnunes | visual symptoms of the study lenses using the |
| | | PRO (MRD) questionnaires. |
| 5.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended |
| | ) | symptoms questionnaire |

| | Visit 5: Treatment 2 Follow-up 2 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 5.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. | |
| 5.7 | Distance and Near<br>Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 5.8 | Visual Performance Distance (4M) Intermediate (64 cm) Near (40 cm) | Binocular Visual performance will be recorded for the following: Distance, Bright Illuminance High and Low Contrast ETDRS Charts 4M-HC#3 and LC#3 Near, Bright Illuminance Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast and Low Contrast Near (40 cm) High Contrast and Low Contrast Note: The room illuminance must be between 7.3 and 7.9 EV (394-597 lux). Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV (181-208 cd/m²). Guillon-Poling, Near Chart Luminance Acceptable Range 10.8- 11.1 EV (223-274 cd/m²). | |
| 5.9 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix H |
| 5.10 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject should not proceed to wear the lenses if any of the following is observed: | |

| | Visit 5: Treatment 2 Follow-up 2 | |
|---|---|---|
| Step | Procedure | Details |
| | | <ul> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> </ul> |
| | | <u>NOTE</u> : If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses, and complete the Final Evaluation forms. |
| 5.11 | Collection of unworn lenses (if applicable) | Collect unworn lenses returned by the subject. |
| 5.12 | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. NOTE: Lenses do not need to be stored in a refrigerator. |
| 5.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 5.14 | Continuance | Determine whether the subject is eligible to continue in the study based on the examination findings. |

| | Visit 5: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 5.15 | Lens Selection | Select the same lens pair and power that was dispensed at Visit 4. Record the Test lens parameters (power and lot number). |
| 5.16 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated from the other worn lenses that will be |

| | Visit 5: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| | | shipped back to the Sponsor. Complete the |
| | | Product Quality Complaint form. |
| 5.17 | Lens Settling | Allow the study lenses to settle for a |
| | | minimum of 10 minutes. |
| 5.18 | Determine Visual | Determine if the subject's vision is acceptable |
| | Satisfaction | with the lenses. Allow the subject to look |
| | | down a hallway or out of a window for |
| | | distance vision assessments, and for them to |
| | | read a book, magazine or similar for near |
| | | vision. |
| 5.19 | Distance and Near | Measure the distance and near visual acuity |
| | Entrance Visual | OD, OS and OU. Record the results. |
| | Acuity | 1 77777 2000 |
| | | For near measures use the ETDRS 2000 |
| | | Series Chart 1 or 2. The acuity will be |
| | | recorded to the nearest letter OD, OS and |
| 5.20 | D: 4 O | OU. |
| 5.20 | Distance Over- | Perform a distance over-refraction OD and |
| | Refraction and | OS using loose lenses outside of the |
| | Distance Visual | phoropter under ambient room illumination. |
| | Acuity | The distance over-refraction may also be refined under binocular conditions. Record |
| | | the results. The results of the distance over- |
| | | refraction may also be checked for the impact on near vision under monocular and/or |
| | | binocular conditions. |
| 5.21 | Lens Fit Assessment | Evaluate overall lens fit acceptance |
| 3.21 | Lens I'it Assessment | (acceptable or unacceptable) based on |
| | | centration, movement and other fitting |
| | | characteristics. |
| | | Characteristics. |
| | | An unacceptable fit is deemed by one of the |
| | | following criteria: |
| | | • limbal exposure at primary gaze or |
| | | with extreme eye movement; |
| | | • edge lift; |
| | | <ul><li>edge int,</li><li>excessive movement in primary and</li></ul> |
| | | up gaze; or |
| | | • insufficient movement in all three of |
| | | the following conditions: primary |
| | | gaze, up gaze, and Josephson push up. |
| | | 5-2-, or 5-2-, and cosephson pash up. |

| | Visit 5: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details Details |
| | | <u>NOTE</u> : If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses, and complete the Final Evaluation forms. |
| 5.22 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. NOTE: The distance visual acuity must be at |
| | | least 20/30 OU for the lenses to be dispensed. |
| 5.23 | Dispensing Criteria | <ul> <li>The following criteria must be met for lenses to be dispensed and if all are not met the subject will be discontinued.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |
| 5.24 | Patient Instructions | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> </ul> |

| | Visit 5: Treatment 3 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| Step | Procedure | <ul> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> <li>Subjects will be instructed to bring their habitual contacts or glasses to the next visit.</li> <li>NOTE: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging</li> </ul> |
| | | should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. |
| 5.25 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 days. NOTE: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

#### VISIT 6

The subjects must present to Visit 6 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 6: Treatment 3 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 6.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 6.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 6.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 6.4 | PRO (MRD)<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, and visual symptoms of the study lenses using the PRO (MRD) questionnaires. |
| 6.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire |
| 6.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 6.7 | Distance and Near<br>Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 6.8 | Visual Performance<br>Distance (4M)<br>Intermediate (64 cm)<br>Near (40 cm) | Binocular Visual performance will be recorded for the following: Distance, Bright Illuminance High and Low Contrast ETDRS Charts 4M-HC#3 and LC#3 Near, Bright Illuminance |

| | Visit 6: Treatment 3 Follow-up 1 | | |
|---|---|---|---|
| Step | Procedure | Details Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast and Low Contrast Near (40 cm) High Contrast and Low Contrast Note: • The room illuminance must be between 7.3 and 7.9 EV (394-597 lux). • Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV (181-208 cd/m²). • Guillon-Poling, Near Chart Luminance Acceptable Range 10.8- 11.1 EV (223-274 cd/m²). | |
| 6.9 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix H |
| 6.10 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). NOTE: If lens fit is unacceptable subject will be discontinued from the study. Remove the lenses, and complete the Final Evaluation forms. Collect unworm lenses returned by the | |
| 6.11 | Collection of unworn lenses (if applicable) | Collect unworn lenses returned by the subject. | |

| | Visit 6: Treatment 3 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 6.12 | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. NOTE: Lenses do not need to be stored in a refrigerator. |
| 6.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the |
| | | study, indicate the reason. |
| F.2 | Exit Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best-corrected distance visual acuity (OD and OS) to the nearest letter. |
| | | <b>Note</b> : This step is not necessary if the subject was exited due to screen failure. |

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.3 | Exit Slit Lamp Biomicroscopy (for subjects that are | FDA Slit Lamp Classification Scale will be used to grade the findings. |
| | discontinued early) | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. This step is not necessary if the subject was exited due to screen failure. |
| | | <b>Note</b> : This step is not necessary if the subject was exited due to screen failure, or if biomicroscopy was performed as part of the final follow-up visit procedures (i.e., immediately prior to the final evaluation). |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected, as appropriate:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate.
- Date and time of the visit and all procedures completed at the unscheduled visit.
- Review of adverse event and concomitant medications.
- Documentation of any test article dispensed or collected from the subject, if applicable.
- Slit lamp findings (using the Slit Lamp Classification Scale).

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Reason for unscheduled visit | Indicate if the <u>only</u> reason for the visit is that the subject requires additional test articles. If the reason is other than resupply of previously dispensed lenses, specify the reason for the visit. |
| U.2 | Chief Complaints (if applicable) | Record the subject's chief complaints for reasons for the unscheduled visit. |
| U.3 | Adverse Events and<br>Concomitant<br>Medications Review<br>(if applicable) | Review any changes to the subject's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. |
| U.4 | Entrance VA (if applicable) | Record the entrance distance visual acuity (OD, OS) to the nearest letter. |
| U.5 | Subjective Sphero-<br>cylindrical<br>Refraction (if<br>applicable) | Perform bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS). |
| U.6 | Slit Lamp<br>Biomicroscopy (if<br>applicable) | FDA Slit Lamp Classification Scale will be used to grade the findings. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| U.7 | Dispensing (if applicable) | If the subject requires additional lenses to complete the wear period and is eligible to do so, provide additional lenses per the dispensing instructions given in the detailed study procedures. |
| U.8 | Exit Visual Acuity (if applicable) | Record the subject's exit distance visual acuity (OD, OS) to the nearest letter. |

NOTE: If the only reason for the unscheduled visit is that the subject requires additional test articles, only the dispensing information needs to be recorded.

#### 7.4. Laboratory Procedures

Not Applicable

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

#### 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent.
- they are eligible.
- completed all study visits

#### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject withdrawal of consent.
- Subject not compliant to protocol
- Subject lost to follow-up.
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant).
- Subject develops significant or serious adverse events necessitating discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE).
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment).
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled).
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study.
- Record the spherocylindrical refraction with best corrected distance visual acuity.
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in section 7.2.
- Collect all unused test article(s) from the subject.
- Make arrangements for subject care, if needed, due to their study participation

Additional subjects will be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications and therapies are medications or therapies that contraindicate contact lens wear. See the Exclusion criteria for specific details.

#### 9.1. Systemic Medications

The following table lists the medications disallowed in this study.

Table 4: Disallowed systemic medications

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Anticholinergics | Irritable bowel syndrome, Parkinson's disease, peptic ulcer, cystitis, nasal congestion, cold symptoms, overactive bladder, COPD | Bentyl, Spiriva, Atrovent,<br>Hyosyne, Levsin, Symax Fastab,<br>Symax SL, Homax SL, Cogentin,<br>Transderm Scop, etc., |
| Oral<br>Phenothiazines | Antipsychotic disorders (schizophrenia, mania) | Compazine, Mellarill, Thorazine, Phenagran, etc |
| Oral Retinoids | Cystic acne | Isotretinoin |
| Corticosteroids | Arthritis, colitis, asthma, bronchitis, allergic or inflammatory conditions | Cortisone, Prednisone,<br>Hydrocortisone, Medrol, Kenalog<br>etc., |
| Oral Tetracycline | Urinary Tract Infection, acne, chlamydia, gonorrhea | Sumcyin, Acitsite, Achromycin V, etc. |

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and as required, to the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study, then it must be reported to IEC/IRB. This is a "Major Deviation". Deviations that contradict the information contained in the Informed Consent/Assent forms will be considered Major Deviations.

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature.

Protocol waivers are prohibited.

Table 5 lists examples of deviations that will constitute major and minor protocol deviations for this study.

Table 5: Examples of major and minor protocol deviations

| Deviation category | Major deviation | Minor deviation |
|---|---|---|
| Out-of-window visit | Visit attended more than 2 days out of visit window defined in study procedures | Visit attended 2 or fewer days out of visit window defined in study procedures |
| Unanswered PRO questions | For questionnaires where data is related to a primary or secondary endpoint, more than 2 PRO questions are unanswered (i.e., left blank). | For questionnaires where data is related to a primary or secondary endpoint, 2 or fewer PRO questions are unanswered (i.e., left blank). For questionnaires where data is not related to a primary or secondary endpoint, any PRO questions are unanswered (i.e., left blank). |

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

#### 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.

- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return (Refer to Form Control No. for test article return instructions).

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also apply and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device."

**Note**: This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices.

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.

**Note**: Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

**Serious Adverse Event (SAE)** – An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.

- Chronic disease
- Foetal distress, foetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)

- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device."

NOTE 1: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

NOTE 2: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device.

**Unanticipated Adverse Device Effect (UADE)** – A UADE is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

#### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related, unlikely related, possibly related, or related see definition in section 13.2.1).
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild, moderate, or severe see definition in section 13.2.2).
- Outcome not recovered or not resolved, recovering or resolving, recovered or resolved with sequelae, recovered or resolved, death related to adverse event, or unknown.
- Actions Taken none, temporarily discontinued, permanently discontinued, or other.

#### 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

• Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.

- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

#### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

#### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs and complete the Adverse Event eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

• Adverse event (diagnosis not symptom).

- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted (where appropriate), including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event, if the AE is related to the visual system.

Upon discovery of an AE that is deemed 'possibly related' or 'related' to the test article or study procedures (whether related to the visual system or not), an AE review form must be completed. Additional dated and initialed entries should be made at follow-up evaluations. Separate forms must be completed for each eye if the AE is bilateral.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1. Reporting Adverse Events to Sponsor

### Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately.
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

#### **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

### 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according to the written guidelines, including reporting timelines.

#### 13.5. Event of Special Interest

None

### 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below. More details will be included in the stand-alone Statistical Analysis Plan (SAP). The SAP will be developed and finalized prior to database lock.

All data summaries and statistical analyses will be performed using the Statistical Analysis System (SAS) software Version 9.4 or higher (SAS Institute, Cary, NC).<sup>15</sup> Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (Descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

Summaries will be presented by separately for each lens type (Test and Control) and time point (baseline, fitting, 3-Day follow-up, 1-week follow-up, exit evaluation and unscheduled visits

(when applicable)) and will be performed separately by completion status (Safety Population, Per-Protocol Population and Intent-to-Treat, when appropriate).

### 14.2. Sample Size Justification

This study was designed and powered to test for superiority of the Test lens relative to the DT1MF lens after 1-week of optimized lens wear with respect to clarity of vision in dim or low lighting and clarity of vision when reading in dim light. Additionally, this study was also powered to test the following after 1-week of optimized lens wear: superiority of the Test lens compared to DT1MF with respect to clarity of intermediate and near vision as well as non-inferiority with respect to clarity of distance vision.

The sample size for co-primary endpoints was estimated to achieve a minimum statistical power of 90% using a 2-sided type I error rate of 5% each and a minimum statistical power of 90% for the secondary endpoints using a 2-sided type I error rate of 1.67% each (5% familywise error rate).

Historical data from two study was utilized in the sample size calculation for this study. Both clinical studies, were 2x3 crossover designs with 1-week follow-up evaluation for the optimized lens wear. Table 6 below summaries the historical studies and Table 7 displays the estimated odds ratio and corresponding 95% CIs.

Table 6: Summary of Historical Studies Included in Sample Size Calculations

| Study<br>Number | Population | Design | Number<br>Enrolled | Number<br>Completed | Number included in PP population | Number in<br>ITT<br>population |
|---|---|---|---|---|---|---|
| Tuilibei | | - 0 | | | | population |
| | Hyperopes | 2x3 | 78 | 75 | 64 | 75 |
| | Myopes | 2x3 | 81 | 78 | 66 | 78 |

PP: Per-Protocol; ITT: Intent-to-treat

Table 7: Historical Odds Ratio Estimates and 95% CIs – Intent-to-Treat Population

| | | <b>Estimated Odds</b> | 95% Confidence |
|---|---|---|---|
| Endpoint Type | Item | Ratio | Interval |
| Primary | Clarity of vision in low | 1.67 | (1.10, 2.53) |
| | lighting conditions | | |
| | Clarity of vision when | 1.88 | (1.26, 2.82) |
| | reading in low light | | |
| Secondary | Clarity of distance vision | 1.27 | (0.82, 1.98) |
| | Clarity of intermediate | 1.98 | (1.25, 3.13) |
| | vision | | |
| | Clarity of near vision | 2.28 | (1.49, 3.48) |

Odds ratios were calculated as Test over DT1MF

Odds ratio represents odds of having a more positive experience while wearing the Test lens compared to DT1MF

#### Primary and Secondary Sample Size Estimates

Sample size estimates for each co-primary and secondary endpoint were carried out separately using an approximation of the power of an F-test derived from the non-centrality parameter calculated from the observed F statistic of a linear model. Each endpoint was analyzed individually using a generalized linear mixed model with a multinomial distribution and the cumulative logit as the link function. Sequence of lens wear, period, lens and first order carryover effect were included in the model as fixed effects. Study nested within site was included as a random effect (G-side). Errors between measurements within the same subject across periods was model using a variance component (VC) covariance structure. The Kenward and Roger method was used for the calculation of the denominator degrees of freedom.<sup>16</sup>

To estimate the sample size for each co-primary and secondary endpoints, the odds ratio and the cumulative log-odds from the model described above for each endpoint was used to create a new dataset with the same structure and design as the historical studies. This new dataset was then analyzed using a generalized linear model with a multinomial distribution and the cumulative logit as the link function. Lens type was included as the only fixed effect; errors between measurements within the same subject across periods was model using a variance component (VC) covariance structure. The Kenward and Roger method was used for the calculation of the denominator degrees of freedom. The statistical power of each endpoint was calculated using the F-statistics as Power=P(F[Fcrit, v, ncp] > Fcrit); where Fcrit is the critical value of the central F distribution (Fcrit= $F_{[numdf,dmdf,0,alpha]}$ ) under Ho (Ho: centrality param = 0), v is the magnitude of the departure from Ho and ncp is the non-centrality parameter (Stroup).<sup>17</sup>

Table 8 displays the sample size estimates and associated power by endpoint. As indicated below, co-primary endpoints were powered  $\sim$ 92% individually yielding a combined power of  $\sim$ 85%. With respect to secondary endpoints, each hypothesis was also powered to at least  $\sim$ 96% power provided a combine power of  $\sim$ 93%. Therefore, the overall combined study power for co-primary and secondary hypotheses is 79.2% and is considered reasonable to support any conclusions from these analyses.

Table 8: Sample Size Estimates by Endpoint

| Endpoint | | | # of Subjects | |
|---|---|---|---|---|
| Type | Item | Alpha | Complete | Power (%) |
| Primary | Clarity of vision in low lighting conditions | 0.05 | 110 | 92 |
| | Clarity of vision when reading in low light | 0.05 | 69 | 92 |
| Secondary | Clarity of distance vision (non-inferiority) | 0.0167 | 83 | 99 |
| | Clarity of intermediate vision | 0.0167 | 110 | 98 |

| Endpoint | | | # of Subjects | |
|----------|------------------------|--------|---------------|-----------|
| Type | Item | Alpha | Complete | Power (%) |
| | Clarity of near vision | 0.0167 | 110 | 96 |

Based on the table above a total of at least 110 subjects are required to complete the study. To account for screen failures and subject dropout up to 130 hyperopic and myopic subjects will be targeted to be enrolled in this study to the aim of 110 (N=66, myopes and N=44 hyperopes) to complete. The allocation of 1:1.5 (hyperopes: myopes) was chosen based on the market representation and availability of subject population.

#### 14.3. Analysis Populations

#### **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

### **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

### **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

#### 14.4. Level of Statistical Significance

Co-primary endpoints will be tested using a 2-sided error rate of 5% each. Both primary hypotheses must be met in order to test the secondary hypothesis. A Bonferroni correction will be utilized for the adjustment of multiple secondary hypotheses using a 2-sided type I familywise error rate of 5%. All primary and secondary hypotheses must be met in order to test any exploratory hypotheses.

Exploratory hypotheses if tested, will utilize all available historical data in addition to data collected from the current study. Exploratory hypotheses will be tested sequentially by group, where all hypotheses in a preceding group must be met in order to continue any exploratory hypothesis testing. Within each grouping, a Bonferroni adjustment will be utilized to adjust for multiple testing.

#### 14.5. Primary Analysis

The primary analyses will be conducted on the intent-to-treat population.

<u>Clarity of Vision in Dim or Low Lighting and Clarity of Vision when Reading in Dim light</u> Subjective responses for co-primary endpoint will be the outcome (*aval*) defined as category one if a subject responds' 'Excellent' or 'Very Good', the outcome is defined as category two

if a subject responds' 'Good' and the outcome is defined as category three if a subject responds' 'Fair' or 'Poor'.

Since both co-primary endpoints assess various aspects of vision in dim or low light, the association between the two endpoints will be assessed using a Cochran-Mantel-Haenszel chi-square test using the Frequency PROCEDURE in SAS 9.4. If the association between the co-primary endpoints is statistically significant at an alpha=0.05 then the following analysis methods will be implemented:

#### Primary Analysis Plan A (If associate between co-primary endpoints is significant)

The outcomes for co-primary endpoints will be analyzed together using a hierarchical generalized linear mixed model (GLMM) with a multinomial distribution and the cumulative logit as the link function. Sequence of lens wear, period, lens type, first order carryover effect, item and the interaction between lens by item will be included as fixed effects. Site and subject nested within site will be included as random effects. Residual errors between measurements within the same subject and period across items will be modeled using an unstructured covariance (UN) structure. If this structure fails to converge then a variance component (VC) structure will be used. The Kenward and Roger method will be used for the calculation of the denominator degrees of freedom.<sup>16</sup>

Comparisons between the Test and DT1MF will be carried separately for each item out using 2-sided 95% confidence intervals (CIs) constructed for the odds ratio (Test over DT1MF). Superiority will be concluded if a lower limit of a 95% CI is above 1.

#### The Model:

Let  $aval_{ijkl} = (aval1_{ijklm}, aval2_{ijklm}, aval3_{ijklm})$  denote the rating for  $l^{th}$  subject at the  $m^{th}$  site assigned to the  $k^{th}$  sequence for the  $i^{th}$  study lens during the  $j^{th}$  study period (i=1, 2; j=1, 2, 3; k=1,2; l=1.... $n_m$ ; m=1,...,10). As previously described possible values of  $aval_{ijklm}$  are  $aval_{ijklm}$ =1 if a subject responds: 'Excellent' or 'Very Good',  $aval_{ijklm}$ =2 if a subject responds: 'Good' and  $aval_{ijklm}$ =3 if a subject responds: 'Fair' or 'Poor'. The Likelihood will be constructed as follows:

$$\begin{aligned} aval_{ijklm} \sim & \text{Multinomial } (p1_{ijklm}, p2_{ijklm}, p3_{ijklm}) \\ & p1_{ijklm} = aval1_{ijklm} \\ & p2_{ijklm} = aval2_{ijklm} - aval1_{ijklm} \\ & p3_{ijklm} = 1 - \sum_{X=1,2} pX_{ijklm} \end{aligned}$$

$$\text{Logit} \left( avalX_{ijklm} \right) = \beta_o + \beta_1 * sequence_k + \beta_2 * period1_j + \beta_3 * period2_j + \beta_4 * \\ lens_{i[j,k]} + \beta_5 * carry_{i[j,k]} + \beta_6 * item_h + \beta_7 * item_h * lens_{i[j,k]} + \delta_m + \gamma_{lm} + \varepsilon_{hijklm}$$

Where,  $\beta_0$  is the intercept for X=1,2,3;  $sequence_k=1$  if Test/DT1MF/DT1MF and  $sequence_k=0$  if DT1MF/Test/Test;  $period1_j=1$  if first period and  $period1_j=0$  otherwise;

;  $period2_j=1$  if second period and  $period2_j=0$  otherwise;  $lens_{i[j,k]}=1$  if Test and  $lens_{i[j,k]}=0$  if DT1MF.  $carry_{i[j,k]}=1$  if lens is Test and  $carry_{i[j,k]}=0$  if lens is DT1MF.

Primary Analysis Plan B (If associate between co-primary endpoints is NOT significant)

The outcome will be analyzed separately for each primary endpoint using a generalized linear mixed model with a multinomial distribution and the cumulative logit as the link function. In each model, sequence of lens wear, period, lens type and first order carryover effect will be included as fixed effects. Site will be included as a random effect. Residual errors between measurements within the same subject across study periods will be modeled using an unstructured covariance (UN) structure. Comparisons between the Test and DT1MF will be carried out using 2-sided 95% confidence intervals (CIs) constructed for the odds ratio (Test over DT1MF). Superiority will be concluded if a lower limit of a 95% CI is above 1.

#### The Model:

Let  $aval_{ijkl} = (aval1_{ijklm}, aval2_{ijklm}, aval3_{ijklm})$  denote the rating for  $l^{th}$  subject at the  $m^{th}$  site assigned to the  $k^{th}$  sequence for the  $i^{th}$  study lens during the  $j^{th}$  study period (i=1, 2; j=1, 2, 3; k=1,2; l=1.... $n_m$ ; m=1,...,10). As previously described possible values of  $aval_{ijklm}$  are  $aval_{ijklm}=1$  if a subject responds: 'Excellent' or 'Very Good',  $aval_{ijklm}=2$  if a subject responds: 'Good' and  $aval_{ijklm}=3$  if a subject responds: 'Fair' or 'Poor'. The Likelihood will be constructed as follows:

$$aval_{ijklm} \sim \text{Multinomial } (p1_{ijklm}, p2_{ijklm}, p3_{ijklm})$$

$$p1_{ijklm} = aval1_{ijklm}$$

$$p2_{ijklm} = aval2_{ijklm} - aval1_{ijklm}$$

$$p3_{ijklm} = 1 - \sum_{X=1,2} pX_{ijklm}$$

$$\text{Logit } (avalX_{ijklm}) = \beta_o + \beta_1 * sequence_k + \beta_2 * period1_j + \beta_3 * period2_j + \beta_4 * lens_{i[j,k]} + \beta_5 * carry_{i[j,k]} + \delta_m + \varepsilon_{ijklm}$$

Where,  $\beta_o$  is the intercept for X=1,2,3;  $sequence_k=1$  if Test/DT1MF/DT1MF and  $sequence_k=0$  if DT1MF/Test/Test;  $period1_j=1$  if first period and  $period1_j=0$  otherwise;  $period2_j=1$  if second period and  $period2_j=0$  otherwise;  $lens_{i[j,k]}=1$  if Test and  $lens_{i[j,k]}=0$  if DT1MF.  $carry_{i[j,k]}=1$  if lens is Test and  $carry_{i[j,k]}=0$  if lens is DT1MF.

## **Hypothesis Testing**

Regardless of which Plan (Primary Analysis Plan A or B) is implemented, superiority testing will be conducted separately for each co-primary endpoint as follows:

Ho:  $OR \le 1$ Ha: OR > 1


Where, the OR represents the odds of having a more positive experience (Excellent or Very Good) while wearing Test compared to DT1MF. Superiority of Test relative to DT1MF will be concluded if a lower limit of a 95% CI is above 1.

#### 14.6. Secondary Analysis

Clarity of intermediate and near vision will be analyzed using the intent-to-treat population while clarity of distance vision will be analyzed using the per-protocol population.

#### Clarity of Distance Vision

Subjective responses to this item (defined as *aval*) will be categorized in the same manner as described for the primary endpoints. The outcome will be analyzed and using the model described for Primary Analysis Plan B above.

### **Hypothesis Testing**

Non-inferiority of the Test compared to DT1MF will be conducted as follows:

Ho:  $OR \le 0.67$ Ha: OR > 0.67

Where, the OR represents the odds of having a more positive experience (Excellent or Very Good) while wearing Test compared to DT1MF. Non-inferiority of Test relative to DT1MF will be concluded if the lower limit of the simultaneous 95% CI (98.33% individually) is above 0.67. A cumulative odds ratio margin of 0.67 was utilized as this corresponds to nomore than a 10% difference using a reference rate of 0.58 for DT1MF.

#### Clarity of Intermediate and Near Vision

Subjective responses to these two items (defined as *aval*) will be categorized in the same manner as described for the primary endpoints. Association between these two endpoints will be assessed using the same test as the primary endpoints and will following the same strategy.

### **Hypothesis Testing**

Regardless of which Plan (Primary Analysis Plan A or B) is implemented, superiority testing will be conducted separately for clarity of intermediate and near vision as follows:

Ho:  $OR \le 1$ Ha: OR > 1

Where, the OR represents the odds of having a more positive experience (Excellent or Very Good) while wearing Test compared to DT1MF. Superiority of Test relative to DT1MF will be concluded if a lower limit of a simultaneous 95% CI (98.33% individually) is above 1.

#### 14.7. Other Exploratory Analysis

If co-primary and all secondary hypotheses are met, then a meta-analysis will be performed on the following exploratory items utilizing data from all historical studies with database hard-

lock (completed after design-lock [Phase 2b]. This will include , , , , , and (if database is hard-locked at the time this analysis is performed). The approximate number of subjects expected from the historical data is 300. The approximate allocation of subjects by study is displayed in Table 9 below.

Table 9 Clinical Studies Planned to be Utilized in Exploratory Meta-Analysis

| Study Number | Population Included | Approximate Allocation of Subjects |
|--------------|----------------------|------------------------------------|
| | Hyperopes | 75 |
| | Myopes | 78 |
| | Hyperopes | 60 |
| | Hyperopes and Myopes | 100 |

is currently in execution; will begin January 2022

Any analyses performed on exploratory endpoints will be on the intent-to-treat population. Statistical analysis will follow the Meta-Analysis approach as discussed in Whitehead <sup>20</sup> This analysis will be discussed completely in the stand-alone SAP.

The stand-alone SAP will include full details describing the following:

- 1. Historical data to be utilized
- 2. Methodology for assessing associations between endpoints within a grouping
- 3. Model details to be utilized for each grouping
- 4. Strategy for adjustments for multiple testing
- 5. Strategies regarding utilizing subject data, if a subject participate in more than 1 historical study
- 6. Methodology for accounting for different study designs

#### 14.8. Interim Analysis

There will not be an interim analysis performed on this study.

#### 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 10%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 50 imputations.

#### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

#### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using the BioClinica EDC system. An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis. External data sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2020.1

#### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication

- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

### 15.3. Trial Registration on ClinicalTrials.gov

This study will be registered on ClinicalTrials.gov based on the following: This study is not an early feasibility study.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

#### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

#### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness

remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

### 16.4. Data Monitoring Committee (DMC)

Not Applicable.

#### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

#### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Subjects will only be enrolled if the subject is fully able to understand the risks, benefits, and potential adverse events of the study and provide their consent voluntarily.

#### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, section 4 of the ICH E6(R2) guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with section 8 of the ICH E6(R2) guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

### 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)

- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH GCP<sup>2</sup> and ISO 14155:2020<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

#### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH GCP guidelines, the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH GCP and all study documents as specified by the applicable regulatory requirement(s).<sup>2</sup> The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated

marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

#### 21. PUBLICATION

There is currently no plan to publish this study in its entirety however the results of the study are intended to be used to support product claims.

#### 22. REFERENCES

- 1. ISO 14155:2020: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at https://www.iso.org/standard/45557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 4. United States (US) Code of Federal Regulations (CFR). Available at https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Karkkainen TR. Investigator Brochure CR-6479 Comparison of a Silicone Hydrogel Daily Disposable Multifocal Contact Lens to a Marketed Product
- 6. Karkkainen TR. Clinical Study Report Evaluation of a Daily Disposable Multifocal Contact Lens with an UV Blocker Additive
- 7. Karkkainen TR. Clinical Study Report Dispensing evaluation of daily disposable multifocal contact lenses in a population of hyperopic presbyopes
- 8. Karkkainen TR. Clinical Study Report Evaluation of a Daily Disposable Novel Multifocal Contact Lens in a Myopic Population
- 9. Karkkainen TR. Clinical Study Report Evaluation of a Daily Disposable Novel Multifocal Contact Lens in a Hyperopic Population
- 10. Karkkainen TR. Clinical Study Report Evaluation of a Daily Disposable Novel Multifocal Contact Lens in a Myopic Population
- 11. Karkkainen TR. Clinical Study Report Evaluation of Investigational Daily Disposable Multifocal Contact Lenses Produced with Different Manufacturing Processes September 08, 2021.
- 12. Karkkainen TR. Clinical Study Report Evaluation of Daily Disposable Multifocal Contact Lenses Made With Two Different Manufacturing Processes September 17, 2021.
- 13. Karkkainen TR. Clinical Study Report Evaluation of Investigational Daily Disposable Multifocal Contact Lenses Produced with Different Manufacturing Processes in Myopes October 11, 2021.
- 14. Karkkainen TR. Clinical Study Protocol Comparison of a Daily Disposable Multifocal Contact Lens to a Marketed Product
- 15. SAS Institute Inc. 2016 SAS/STAT® 14.3 User's Guide. Cary, NC: SAS Institute Inc.
- 16. Kenward MG, Roger JH. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics*. 1997;53(3):983.
- 17. Stroup W. Generalized Mixed Models: Modern Concepts, Methods and Applications. Boca Raton CRC Press; 2013
- 18. Bonferroni C. Calculation of the insurance groups of heads. *Studies in Honour of Professor Salvatore Ortu Carboni*. 1935;Rome: Italy:13-60.
- 19. Karkkainen TR. Clinical Study Protocol Evaluation of a daily disposable silicone hydrogel multifocal contact lens in myopes and hyperopes

- 20. Whitehead A. *Meta-Analysis Of Controlled Clinical Trials*. John Wiley & Sons, Ltd; 2002.
- 21. Health Information Portability and Accountability Act (HIPAA). Available at https://www.hhs.gov/hipaa/for-professionals/privacy/index.html
- 22. Regulation (EU) 2017/745 of the European Parliament and of the Council of 5 April 2017 on medical devices. Available at http://data.europa.eu/eli/reg/2017/745/2017-05-05

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)



CR-6479, v 3.0

5

## APPENDIX B: PATIENT INSTRUCTION GUIDE

A patient instruction guide (PIG) will be provided separately

APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)



a Novartis company

# DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) Soft

Contact Lenses for Daily Disposable Wear

W900038292

IMPORTANT: This package insert is effective as of March 2016 and applicable to the delettion A contact lenses described below. Please read carefully and keep this information for future use. This package insert is intended for the eye care professional, but should be made available to patients upon request. The eye care professional should provide the patient with appropriate instructions that perial to the patient's prescribed lenses. Copies of this package insert are available without charge from Alcon by calling Customer Service at 1-800-241-5999 or download from our website at www.sicon.com. In addition, a Patient instruction Booklet is available which is recommended to be given to patients.



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional.

#### PRODUCT DESCRIPTION

DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (deleflicon A) soft contact lenses are made from a lens material that is 33% water and 67% (deletticon A) polymer, a stilcone containing hydrogel with added phosphatidylcholine. The core lens material containing 33% water transitions through a water gradient to a hydrogel surface layer that exceeds 80% water. Lenses contain the color additive copper phthalocyanine, a light blue tint, which makes them easier to see when handling.

#### Lens Properties

· Refractive Index hydrated: 1.42

93% (@ 610 nm, -1.00D) Light Transmittance: · Oxygen Permeability (Dk): 140 x 10<sup>-11</sup> (cm<sup>2</sup>/sec)(ml

> 02 /ml x mm Hg), measured at 35° C (intrinsic Dk-Coulometric

method)

· Water Content: 33% by weight in normal

saline

· Surface Water Content: > 80%

Lens Parameters

 Diameter Range 13,0 to 15.0 mm · Spherical Power Range -20.00 to +20.00D · Base Curve Range 8.0 to 9.2 mm

#### Lens Parameters Available<sup>3</sup>

#### DAILIES TOTAL1\* (deletilcon A) spherical

· Chord Diameter: 14.1 mm

0.09 mm @ -3.00D (varies Center Thickness:

with power) · Base Curve: 8.5 mm

-0.50 to -6.00D (0.25D Powers:

steps); -6.50 to -12.00D (0.50D steps) +0.50 to +6.00D (0.25D steps)

#### DAILIES TOTAL1\* Multifocal (deleflicon A)

 Chord Diameter: 14.1 mm

0.09 mm @ -3.00D (varies Center Thickness:

with power)

 Base Curve: 8.5 mm

· Powers: +6.00D to -10.00D (0.25D

steps) ADD: LO, MED, HI

NOTE: Hereafter, DAILIES TOTAL1\* spherical lenses and DAILIES TOTAL1\* Multifocal contact lenses will simply be referred to as delefilcon A contact lenses unless product distinction is necessary.

When hydrated and placed on the cornea, deletiicon A contact lenses act as a refracting medium to focus light rays on the retina.

#### INDICATIONS (USES)

DAILIES TOTAL1\* (delefilion A) spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia. and hyperopia) in phakic or aphakic persons with non-diseased eves with up to approximately 1,50 diopters (D) of astigmatism that does not interfere with visual acuity.

DAILIES TOTAL1\* Multifocal (deleflicon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia. and hyperopia) and/or presbyopia in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 (D) or less and who may have up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual

The lenses are to be prescribed for single use, daily disposable wear. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

#### CONTRAIND(CRTKOMB)(REAS(INS NOT TO USE) DO NOT use deleflicon A contact lenses when any of the following exists:

. Inflammation or infection of the anterior chamber of the eye

- Active disease, injury or abnormality affecting the cornea, conjunctiva, or eyelids
- Microbial Infection of the eye
- insufficiency of lacrimal secretion (dry eye) that interferes with contact lens wear
- Corneal hypoesthesia (reduced corneal sensitivity)
- Use of any medication that is contraindicated or interferes with contact lens wear, including eye medications
- Any systemic disease which may be exacerbated by or Interferes with contact lens wear
- · Allergic reactions or ocular irritation of the ocular surfaces or adnexa that may be caused by or exaggerated by the wearing of contact lenses
- Patient history of recurring eye or eyelid infections, adverse effects associated with contact lens wear, intolerance or abnormal ocular response to contact lens wear
- If eyes become red or irritated

#### WARNINGS

Advise patients of the following warnings pertaining to contact lens wear:

- · Problems with contact lenses and lens care products could result in serious injury to the eye. It is essential that patients follow their eye care professional's directions and all labeling instructions for proper use of lenses and lens care products. Serious eye problems, including corneal ulcers, can develop rapidly and lead to loss of vision.
- Daily wear lenses are not indicated for overnight wear, and patients should be instructed not to wear lenses while sleeping. Clinical study results have shown that the risk of serious adverse reactions is increased when contact lenses are worn overnight2.
- Studies2 have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- If a patient experiences eye discomfort, foreign body sensation, excessive tearing, vision changes, or redness of the eye, the patient should be instructed to immediately remove lenses and promptly contact his or her eye care professional. It is recommended that contact lens wearers see their eye care professional regularly as directed.

#### PRECAUTIONS

To prevent damage to the eyes or to the contact lenses, the following precautions should be taken:

Special Precautions for the Eye Care Professional: Due to the small number of patients enrolled in the clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently when selecting an appropriate iens design and parameters, the eye care professional should consider all characteristics of the lens that can affect lens performance and ocular health, including coygen permeability, central and peripheral thickness and optic zone diameter. The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore the continuing ocular health of the patient and iens performance on the eye should be carefully evaluated on initial dispensing and monitored on an ongoing basis by the prescribing eye care professional.

- Fluorescein, a yellow dye, should not be used while the lenses are on the patient's eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used, the eyes should be flushed thoroughly with sterile saline solution that is recommended for in eye use prior to inserting lenses. Avoid dispensing saline from an aerosol can directly into the eye.
- Patients who wear contact lenses to correct presbyopia may not achieve the best possible corrected visual aculty for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Before leaving the eye care professional's office, the patient should be able to promptly remove their lenses or should have someone else available who can remove their lenses for them.
- Eye care professionals should instruct the patient to remove the lenses immediately if the eye becomes red or initiated.
- sary to help assure the Routine eye exar continued health of the patient's eyes. Eye care professionals should make arrangereen(12 w/th/2002 patient for appropriate

follow-up visits. Alcon recommends that patients see their eye care professional once each year, or more often, as recommended by the eye care professional.

- Diabetics may have reduced corneal sensitivity and thus are more prone to corneal injury and do not heal as quickly or completely as non-diabetics.
- . Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly.

Eye Care Professionals should carefully instruct patients about the following safety precautions: Handling Precautions:

- . Be sure that before leaving the eye care professional's office the patient is able to promptly remove lenses or have someone else available to remove them.
- · Good hygiene habits help promote safe and comfortable lens wear. Always wash, rinse and thoroughly dry hands with a lint-free towel before handling lenses.
- REMOVE A LENS IMMEDIATELY If an eye becomes red or irritated.
- · Always handle lenses carefully. Never use tweezers or other sharp objects such as fingernalis to remove lenses from the lens container unless specifically indicated for that use.
- . Do not use if blister package is damaged or not sealed completely. This may result in product contamination which can lead to a serious eye infection.
- . Ensure that the correct lens for each eye is available. Shake the blister pack gently prior to opening. Remove the lens from the blister pack by carefully pouring the lens onto the paim of your clean hand. Ensure the lens is right side out. Inspect lenses prior to insertion. Do not insert damaged lenses.
- To insert lenses:
  - Wash and rinse hands thoroughly and dry completely with a clean, lint free towel before handling lenses.
  - Place a lens on the tip of your clean and dry right or left index finger, place the middle finger of the same hand close to lower evelashes and pull down the lower evelid.
  - Use the fingers of the other hand to lift the upper evelid.
  - Place the lens directly on the eye (comea) and gently roll finger away from the lens.
  - Look down and slowly remove the hand, releasing the lower IId.
  - Look straight ahead and slowly remove the other hand, releasing the upper lid.
  - Blink gently.
- . To remove lenses:
  - Wash and rinse hands thoroughly and dry completely with a clean, lint free towel before handling lenses. Make sure hands are clean and completely dry.
  - Blink fully several times.
  - While looking up, slide the lens down onto the white part of the eve
  - Remove the lens by pinching gently between the thumb and forefinger. Do not pinch the eye tissue.
  - If the lens is difficult to grasp, dry fingers once more and try again. Do not use rewetting drops in this instance.
- . If a lens decenters on the eye, it may be possible to recenter it by:
  - Closing the eye and massaging the lens into place, or
  - Looking in the direction of the lens and blinking gently, or - Gently pushing the off-centered lens onto the comea with
  - light finger pressure on the edge of the upper or lower eyelld.
- If a lens tears in the eye it will feel uncomfortable. Advise wearers it is impossible to lose a contact lens or part of a contact iens behind the eye and to remain calm. Lens pieces may be removed by pinching them as for normal lens removal, carefully avoiding pinching the eye tissue. If the lens pieces do not seem to remove easily, rinsing with saline is recommended. If this does not help, the wearer should contact an eye care professional for assistance.

#### Lens Wearing Precautions:

- · Patients should never exceed the prescribed wearing schedule regardless of how comfortable the lenses feel. Doing so may increase the risk of adverse effects.
- · The lens should move freely on the eye at all times. If the lens sticks (stops.jvj.w/iOg/CO/IN/FN/D/E/IN/DN/IN/ANL/recommended directions in the Care for a Sticking Lens section. If non-movement of the lens continues, the patient should be instructed to consult their eye care professional immediately.

- The eye care professional should be consulted about wearing lenses during water sports and water related activities. Exposure to water or other non-sterile liquids while wearing contact lenses in activities such as swimming, water skiling, and hot tubs may increase the risk of ocular infection, including but not limited to Acanthamoeba keratitis.
- Never allow contact lenses to come into contact with non-sterile liquids (including tap water and saliva) as microbial contamination can occur, which may lead to permanent eye
- Eye Irritation, Infection, or lens damage may result if cosmetics, lotion, scap, cream, hair spray, deodorant, aerosol products or foreign particles come in contact with lenses.
- Environmental tumes, smoke, and vapors should be avoided in order to reduce the chance of lens contamination or physical trauma to the cornea.
- Lenses should be disposed of each day upon removal from the
- Discard any lens which has become dehydrated or damaged. Replace with a sterile, fresh, new lens.
- Note the correct lens power for each eye to prevent getting them mixed up.
- Always carry spare lenses with you or have back-up spectacles available.
- Do not share lenses with anyone as this may spread micro-organisms which could result in serious eye health problems.
- Do not use lenses beyond their expiration date.

- Other Topics to Discuss with Patients:
   Periodic eye examinations are extremely important for contact lens wearers. Schedule and conduct appropriate follow-up examinations to determine ocular response. Alcon recommends that patients see their eye care professional once each year or as recommended by the eye care professional.
- Certain medications may cause dryness of the eye, increased lens awareness, lens intolerance, and blurred vision or visual changes. These include, but are not limited to, antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness. Caution patients using such medications accordingly and prescribe proper remedial measures.
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients

Who Should Know that the Patient is Wearing Contact Lenses:

- Patients should inform their health care practitioners that they are wearing contact lenses.
- Patients should inform their employers that they are wearing contact lenses. Some jobs may require the use of eye protection equipment or may require that contact lenses not be

It is strongly recommended that patients be provided with a copy of the DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal Contact Lenses (deleticon A) Patient Instruction Booklet available from Alcon and understand its contents prior to dispensing the lenses.

#### ADVERSE EFFECTS

Patients should be instructed to check eyes regularly to make sure they look well, feel comfortable and vision is clear. Potentially serious complications are usually accompanied by one or more of the following signs or symptoms:

- Moderate to severe eye pain not relieved by removing the lens
- Foreign body sensation
- Excessive watering or other eye secretions including mucopurulent discharge
- Redness of the eyes
- Photophobia (light sensitivity)
- Burning, stinging or itching or other pain associated with the
- Comfort is less compared to when the lens was first placed on
- Poor visual aculty (reduced sharpness of vision)
- Blurred vision, rainbows or halos around objects
- Feeling of dryness

#### WHAT TO DO IF A PROBLEM OCCURS

Patients should be instructed that if any of the above signs or symptoms are noticed, he or she should:

- IMMEDIATELY REMOVE THE LENSES.
- If the discomfort or problem stops, discard the lens and replace it with a new one.
- If the discomfort or problem continues after removing iens(es) or upon insertion of a new iens, IMMEDIATELY remove the lens(es) and contact the eye care professional for identification of the problem and prompt treatment to
- avoid serious eye damage. The patient should be informed that a serious condition such as corneal uicer, infection, corneal vascularization, or

- iritis may be present, and may progress rapidly. Less serious reactions such as abrasions, inflitrates, and bacterial conjunctivitis must be managed and treated carefully to avoid more serious complications.
- Additionally, contact lens wear may be associated with ocular changes that require consideration of discontinuation or restriction of wear. These include but are not limited to local or generalized comeal edema, epithelial microcysts, epithelial staining, inflitrates, neovascularization, endothelial polymegathism, tarsal papillary changes, conjunctival injection

#### ADVERSE EFFECT REPORTING

If a patient experiences any serious adverse effects associated with the use of DAILIES TOTAL1\* brand (deletiicon A) contact lenses, please notify: Alcon Medical Safety in the USA at 1-800-757-9780.

#### FITTING GUIDE AND PATIENT BOOKLET

Conventional methods of fitting contact lenses apply to delefficon A contact lenses. For a detailed description of the fitting techniques, refer to the DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal Contact Lenses (delefficon A) Professional Fitting and Information Guide. Both the professional fitting guide and a patient instruction booklet are available free of charge from:

Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX, USA 76134-2099 1-800-241-5999

#### LENS WEAR & REPLACEMENT SCHEDULES

DAILY WEAR (less than 24 hours, while awake):

- . To avoid tendency of the daily wear patient to overwear the lenses initially, stress the importance of adhering to a proper, Initial wearing schedule. Normal daily wear of lenses assumes a minimum of 6 hours of non lens wear per 24 hour period.
- It may be advisable for patients who have never worn contact lenses previously to be given a wearing schedule that gradually increases wearing time over a few days. This allows more gradual adaptation of the ocular tissues to contact lens wear.
  - · The maximum daily wearing time should be determined by the eye care professional based upon the patient's physiological eye condition because Individual responses to contact lenses vary. There may be a tendency for patients to overwear the lenses initially. The eye care professional should stress the Importance of adhering to the initial maximum wearing schedule. Studies have not been conducted to show that deletiicon A contact lenses are safe to wear during sleep, therefore patients should be advised to remove their lenses while sleeping. Normal daily wear of lenses assumes a minimum of 6 hours of non-lens wear per 24 hour period. Optimum individual wearing schedule will vary.
- Delefficon A contact lenses are intended to be worn once (daily) disposable wear) and then discarded at the end of each wearing period. The patient should be instructed to start the next wearing period with a fresh new lens.

#### EMERGENCY LENS CARE

Cleaning and disinfection of daily disposable lenses is not recommended. The patient should be reminded to have replacement lenses or back-up spectacles available at all times.

#### CARE FOR A STICKING LENS

If the lens sticks (stops moving) or begins to dry on the eye, instruct the patient to apply several drops of a recommended lubricating solution (used in accordance with package labeling). The patient should walt until the lens begins to move freely on the eye before attempting to remove it. It is important that the patient wash and dry their hands thoroughly before removing the lens. If the lens continues to stick, the patient should IMMEDIATELY consult the eye care professional.

#### IN OFFICE USE OF TRIAL LENSES

Eye care professionals should educate contact lens technicians concerning proper use of trial lenses.

Each contact lens is shipped sterile in a blister pack containing phosphate buffered saline solution. Hands should be thoroughly washed and rinsed and dried with a lint-free towel prior to handling a lens. In order to ensure sterlity, the blister pack should not be opened until immediately prior to use. For fitting and diagnostic purposes lenses should be disposed of after a single use and not be re-used from patient to patient.

#### EMERGENCIES

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should:

Flush eyes Immodiately with tap water or fresh saline solution and in the eye care professional or visit a hospital emergency room without delay.

#### HOW SUPPLIED

Each lens is packaged in a foll-sealed plastic container containing phosphate buffered saline solution with approximately 0.3% of polymeric wetting agents consisting of copolymers of polyamidoamine and poly(acrylamide-acrylic) acid and is steam sterilized seeks] . The package is marked with the base curve, diameter, dioptric power and ADD power (multifocal lenses), manufacturing lot number and expiration date.

The following may appear on the labels or cartons:

| Symbols/Signs/<br>Abbreviations | Description |
|---|---|
| Renty | CAUTION: Federal law (United States) restricts this device to sale by or on<br>the order of a licensed eye care professional. |
| STURBLE | Steam sterflized |
| ≅ EXP | Use by date (Expiry date) |
| LOT | Batch code |
| 2 | Do not reuse |
| (S) | Do not use if blister package is damaged |
| en | Example of two letter language code (English) |
| DIA | Diameter |
| BC | Base curve |
| PWR | Power |
| D | Diopter (lens power) |
| ADD | Addition power |
| C€œs | European conformity sign |
| | Caution |
| T3 | See product instructions |
| 80 NP | Authorized Representative European Community |
| | Manufacturer |
| 0 | Packaging waste license sign |

a trademark of Novartis © 2016 Novartis

Manufacturer: Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX, USA 76134-2099 www.alcon.com 1-800-241-5999

March 2016

w900038292-0316

- 1 Check for actual product availability as additional parameters may be Introduced over time
- <sup>2</sup> Schein, OD, Glynn RJ, Poggio EC, Seddon JM, Kenyon KR. The Relative Risk of Ulcerative Keratitis Among Users of Daily Wear and Extended Wear Soft Contact lenses. N Eng J Med. 1969; 32321 (12):773-783







## APPENDIX E: OCULAR DOMINANCE



## APPENDIX F: LENS FITTING GUIDE





APPENDIX G: CONTROL LENS FITTING GUIDE
# Professional Fitting and Information Guide

DAILIES TOTAL1®
and
DAILIES TOTAL1® Multifocal
(delefilcon A) Soft Contact Lenses
For Single-Use, Daily Disposable Wear

**Water Gradient One-Day Contact Lenses** 



Caution: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional.

°R\_6479\_v 3.0



This page intentionally left blank

#### **Table of Contents**

| | ilon | |
|-----------|-------------------------------------------------|-----|
| Product | Description | 5 |
| | Lens Properties | |
| | Available Lens Parameters | |
| | ns (Uses) | |
| | cations, Warnings, Precautions, Adverse Effects | |
| Adverse | Effect Reporting | 7 |
| Fitting G | uidelines (Spherical Lenses) | |
| | Patient Selection | |
| | Pre-fitting Examination | |
| | Trial Lens Evaluation | |
| | Lens Base Curve Selection | |
| | Initial Lens Power Selection | |
| | Lens Fit Assessment | |
| | Final Lens Power Determination | |
| Fitting G | uidelines (Multifocal Lenses) | .11 |
| | Pre-Fitting Examination | |
| | Patient Selection | |
| | Initial Lens Selection | |
| | Initial Lens Fitting Evaluation | |
| | Initial Lens Visual Evaluation | |
| | Fitting Procedures | |
| Fitting G | uidelines (Monovision) | |
| | Patient Selection | |
| | Eye Selection | |
| | Special Fitting Considerations | |
| | Near Add Determination | |
| | Trial Lens Fitting | |
| | Adaptation | |
| | Other Suggestions | |
| Dispensi | ng Visit | |
| | Follow-Up Examinations | |
| | Follow-up Examination Procedures | |
| Lens Ha | ndling Hints | |
| | Lens Insertion | |
| | Lens Removal | |
| | Care for a Sticking Lens | |
| | Care of Trial Lenses | |
| | and Recycling | |
| | al Information | |
| | Package Insert | |
| Vertex D | istance Conversion Chart | 28 |

This page intentionally left blank

#### INTRODUCTION

Thank you for prescribing DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) daily disposable soft contact lenses. The benefits of a high oxygen transmissible and wettable lens material with a state of the art manufacturing process are combined to make DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) lenses. This guide contains important information regarding fitting procedures and aftercare of the DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) contact lens patient.

#### **Daily Disposability**

By eliminating the need for lens care, daily disposable lenses offer your patients a major advancement in wearing convenience. The next time you prescribe lenses consider the health and comfort benefits of beginning each wearing period with a new pair of fresh, sterile lenses that are worn once and then discarded.

#### LightStream® Lens Technology

DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) contact lenses are made from a proprietary silicone hydrogel material with a water content of approximately 33% water. The use of process automation, precision glass and quartz molds and photolithographic edge forming help ensure every lens has the same crisp optics, smooth surface finish and consistent edge quality from lens to lens. Delefilcon A contact lenses are produced under strictly controlled process conditions and inspected to exacting quality tolerances. As a result, you can be confident your patients will experience consistent vision, comfort, and ease of handling every day.

#### PRODUCT DESCRIPTION

DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal soft contact lenses are made of a silicone containing hydrogel that is approximately 33% water and 67% delefilcon A polymer with added phosphatidylcholine. The core lens material containing 33% water transitions through a water gradient to a hydrogel surface layer that exceeds 80% water. This structure enables a silicone hydrogel lens with a water gradient that has:

- Over 80% water at the surface of the lens to mimic the water content of the cornea.
- · High level of oxygen transmissibility through the lens.
- Excellent overall comfort.

The lenses contain and release phosphatidylcholine (DMPC), a phospholipid found naturally in the tears. In addition, lenses contain the color additive copper phthalocyanine, a light blue tint which makes them easier to see when handling.

The lenses are packaged in strips of 5 individual blisters containing buffered saline with approximately 0.3% of polymeric wetting agents consisting of copolymers of polyamidoamine and poly(acrylamide-acrylic acid).


#### **Lens Properties**

• Refractive Index (hydrated): 1.42

Light Transmittance: ≥ 93% (@610 nm, -1.00D)
 Oxygen Permeability (Dk): 140 x 10<sup>-11</sup> (cm²/sec)

(ml O<sub>2</sub>/ml x mm Hg), measured at 35°C, (intrinsic Dk - Coulometric method)

• Water Content: 33% by weight in normal saline

• Surface Water Content: ≥ 80%

#### Available Lens Parameters<sup>1</sup>

#### DAILIES TOTAL1® (delefilcon A) spherical contact lenses

• Chord Diameter: 14.1 mm

Center Thickness: 0.09 mm @ -3.00 D (varies with power)

Base Curve: 8.5 mm

Powers Available: -0.50 to -6.00 D (0.25 D steps);

-6.50 to-12.00 D (0.50 D steps) +0.50 to +6.00 D (0.25 D steps)

#### DAILIES TOTAL1® Multifocal (delefilcon A) contact lenses

• Chord Diameter: 14.1 mm

• Center Thickness: 0.09 mm @ -3.00 D (varies with power)

Base Curve: 8.5 mm

• Powers: -0.25 to -10.00 D (0.25 D steps);

plano to +6.00 D (0.25 D steps)

ADD: LO, MED, HI

<sup>1</sup>Check for actual product availability as additional parameters may be introduced over time.

#### **ACTIONS**

When hydrated and placed on the cornea delefilcon A soft contact lenses act as a refracting medium to focus light rays on the retina.

#### **INDICATIONS (USES)**

**DAILIES TOTAL1**® (delefilcon A) spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

**DAILIES TOTAL1® Multifocal** (delefilcon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) and/or presbyopia in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 (D) or less and who may have up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

The lenses are to be prescribed for single use, daily disposable wear. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

See WARNINGS for information about the relationship between wearing schedule and corneal complications.

# CONTRAINDICATIONS, WARNINGS, PRECAUTIONS AND ADVERSE EFFECTS

For additional important prescribing and safety information, refer to the Package Insert that is printed in the back of this guide.

#### **ADVERSE EFFECT REPORTING**

If a patient experiences any serious adverse effects associated with the use of DAILIES TOTAL1® or DAILIES TOTAL1® Multifocal (delefilcon A) contact lenses, in the USA please **contact Alcon Medical Safety at** 1-800-757-9780.

#### **FITTING GUIDELINES**

Please see the appropriate sections of this booklet that contain guidelines for spherical, multifocal and monovision fitting techniques.

#### FITTING GUIDELINES (Spherical Lenses)

#### 1. Patient Selection

The patient characteristics necessary to achieve success with DAILIES TOTAL1® (delefilcon A) spherical lenses are similar to those for other spherical soft contact lenses. A thorough pre-fitting examination should be conducted to ensure the patient is a suitable candidate for soft contact lens wear.

The following procedures should be followed when fitting DAILIES TOTAL1® (delefilcon A) spherical lenses. For additional tips on fitting the monovision patient refer to the section *Monovision Fitting Guidelines*.

#### 2. Pre-fitting Examination

#### A pre-fitting examination is necessary to:

- assess the patient's motivation, physical state and willingness to comply with instructions regarding hygiene and wear schedule
- make ocular measurements for initial contact lens parameter selection
- collect baseline clinical information to which post-fitting examination results can be compared

#### A pre-fitting examination should include:

- · a thorough case history
- · a spherocylindrical refraction
- keratometry
- · tear film assessment
- biomicroscopy

#### 3. Trial Lens Evaluation

#### A. Lens Base Curve Selection

A well-fitted lens provides good movement, centration and comfort. An optimal fit can be achieved for the vast majority of patients with the single 8.5 mm base curve.

#### B. Initial Lens Power Selection

The initial power selection should be as close as possible to the patient's prescription after taking into account spherical equivalent and vertex calculations, if necessary.

#### **Spherical Equivalent Calculation**

To determine initial lens power, convert the spherocylindrical spectacle Rx to its spherical equivalent as follows:

Spherical Equivalent = Sphere power + 1/2 (Cylinder Power)
Example: Spectacle Rx: -4.50D -1.00 x 180

Spherical equivalent: -4.50D + (-0.50D) = -5.00D

#### **Vertex Distance Conversion**

If the spherical equivalent is greater than  $\pm$  4.00D, a vertex distance correction is necessary (see *Vertex Distance Conversion Chart*) to determine the lens power required at the corneal plane.

Example: Spectacle Rx: -4.50D -1.00 x 180

Spherical equivalent: -4.50D + (-0.50D) = -5.00D Vertex compensation: -4.75 (initial lens power)

CR-6479, v 3.0




#### C. Lens Fit Assessment

Allow the lenses to settle on the eyes for approximately 10 minutes. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate.

Evaluate the fit and movement of the lenses on the eye in primary and up gaze positions. The **Push-up Test**, as described below, is an additional test of the lens evaluation. The following guidelines will be helpful in fit evaluation:

#### Characteristics of a Well-fitted Lens

A well-fitted DAILIES TOTAL1® (delefilcon A) spherical contact lens satisfies the following criteria:

- 1. Good centration and full corneal coverage in all fields of gaze.
- Sufficient lens movement to allow tear exchange under the lens during a blink in primary or upward gaze.
- 3. Satisfactory Push-up Test
  - This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then pull the lid back down and observe the return of the lens.
  - A well fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- Good comfort and stable visual response (with over refraction).

#### Characteristics of a Tight (Steep) Lens Fit

A tight or steep lens fit would display some or all of the following characteristics:

- Insufficient or no lens movement during a blink in primary or upward gaze.
- 2. Unsatisfactory Push-up Test
  - A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- 3. Good centration.
- 4. Good comfort.
- 5. Fluctuating vision between blinks.

#### Characteristics of a Loose (Flat) Lens Fit

A loose lens fit would display some or all of the following characteristics:

- 1. Reduced comfort, usually accompanied by lower lid sensation.
- Poor centration with limbal exposure on exaggerated eye movement.
- 3. Lens edge standoff.
- 4. **Excessive lens movement** during the blink in primary or upward gaze.
- 5. Unsatisfactory Push-up Test
  - A loose fitting lens will move easily but may remain decentered or slip under the upper lid.



An inverted lens may mimic the characteristics of a loose lens. If any of the above signs occur remove the lens and check to make sure it is not inverted.

#### **General Fitting Tips**

- Trial fitting of the individual eye is recommended.
- A well-fitted lens will show movement of 0.1 to 0.5 mm.

#### D. Final Lens Power Determination

After the characteristics of a well fitted lens have been satisfied, conduct a **spherical over-refraction** to determine the proper lens power to be dispensed.

Example: Diagnostic lens: -4.50

Over-refraction: -0.25 Final lens power: -4.75

#### FITTING GUIDELINES (Multifocal)

The **DAILIES TOTAL1® Multifocal** (delefilcon A) soft contact lens is a progressive aspheric simultaneous vision soft contact lens, intended to correct presbyopia with or without additional ammetropia, available in three ADD powers; low (LO), medium (MED) and high (HI). For each lens the near and intermediate powers are concentrated primarily in the central portion of the optical zone while the distance power is contained in the surrounding portion. The continuous changes in power across the surface of the lens allow patients requiring a reading addition of up to + 3.00D to see clearly at far, intermediate, and near distances.

Achieving high success with DAILIES TOTAL1® Multifocal (delefilcon A) contact lenses is dependent on several factors, including the patient's motivation, expectations and visual wearing environment, as well as your skill in optimizing the lens powers to balance binocular performance at distance and near. The information in this guide is designed to provide you with the tools to manage your presbyopic patients through each stage of the process from the initial case history to post-fitting follow-up.

#### 1. Pre-fitting Examination

#### A pre-fitting examination is necessary to:

- determine whether a patient is a suitable candidate for DAILIES TOTAL1® Multifocal (delefilcon A) contact lenses
- make ocular measurements and assessments for initial contact lens parameter selection
- collect baseline clinical information to which post-fitting examination results can be compared

#### A pre-fitting examination should include:

- a thorough case history
- detailed assessment of patient's individual visual demands
- understanding of patient's objectives for lens wear and expectations
- a distance spherocylindrical refraction, near add determination and measurement of pupil diameter
- keratometry
- tear assessment
- biomicroscopy

Note: The importance of a thorough case history should not be underestimated. The information gained through careful listening and probing will help greatly in satisfying each patient's unique needs.

#### 2. Patient Selection

The eye care professional should weigh several factors when considering patient selection for a DAILIES TOTAL1® Multifocal (delefilcon A) soft contact lens fitting. When fitting a lens intended to correct for presbyopia, it is especially important to evaluate the particular visual needs, objectives, lifestyle and expectations of the individual patient. Prospective candidates may include current contact lens wearers, former wearers, and persons with no previous wear history. For former wearers it is important to determine the cause for discontinuation.

There are two general categories of candidates based on anticipated usage: those who seek to wear their lenses as their principal means CR-6479, v 3.0


of vision correction, and those who wish to integrate the use of their contact lenses with spectacles. The integrative user often seeks to wear their lenses for sports or other occasional activities while reverting to spectacles under poor lighting or otherwise demanding vision conditions. In general, even the part-time user does not require more than a few moments re-adaptation time following an interval of no lens wear.

While candidates with greater than 1.00 diopter of refractive error have often been thought of as better candidates than those with low error or emmetropia, this is a generalization that often does not hold true for a given individual. Success is influenced by many factors and the eye care professional is encouraged to offer DAILIES TOTAL1® Multifocal (delefilcon A) contact lenses to all interested presbyopic patients who satisfy the standard requirements for soft contact lens wear.

To summarize patient selection, the characteristics of "ideal candidates" and those that will be more difficult to fit" are listed below:

#### Ideal Candidates

- Refractive cylinder < 1.00D.</li>
- Attainable visual demands that do not depend upon resolving very fine (smaller than 20/20 letters) details at both distance and near for extended periods while wearing DAILIES TOTAL1® Multifocal contact lenses.
- Emphasis on tasks where it is advantageous to have objects simultaneously in focus over a large range of viewing distances.
- Expectations consistent with actual everyday visual demands.
- Motivated to wear lenses and understands that vision may not always be as sharp as with spectacles for some distances or lighting conditions.
- Unable to adapt to monovision correction.

#### Less than Ideal Candidates

- Critical or very fine visual demands at both distance and near.
- Refractive cylinder ≥ 1.00D (any axis) in one or both eyes or against-the-rule refractive cylinder > 1.00D in one or both eyes.
- Monocular distance acuities poorer than 20/20 with spherical equivalent refractive correction.
- Myopic anisometropia where the refractive error for one of the two eyes is low (≤1.50D) and has not been habitually corrected.
- Pupil size larger (> 4 mm) or smaller (<3 mm) than norm for presbyopic population under natural illumination conditions.
- Abnormal binocular sensory function (e.g., amblyopia or strabismus).
- Expectation to discard and never use spectacles again, including reading glasses, even for special tasks or viewing conditions.
- Highly satisfied monovision wearers.
- Any other contraindications to successful contact lens wear such as tear abnormality or lid margin disease.

#### 3. Initial Lens Selection

#### A. Initial Base Curve Selection

DAILIES TOTAL1® Multifocal (delefilcon A) contact lenses are available in a single 8.5 mm base curve.

#### **B. Initial Lens Power Selection**

Note: A careful maximum plus spherocylindrical refraction and near-point add determination should be conducted prior to selecting a DAILIES TOTAL1® Multifocal (delefilcon A) trial lens. Auto-refraction findings should be refined manually to rule out effects of instrument myopia and ensure proper control of residual accommodation.

The DAILIES TOTAL1® Multifocal lens design makes selecting the initial lens power easy. You need only manipulate the distance power. The optimum starting point is with a power that is equal to or *more plus or less minus* than the vertex corrected spherical equivalent spectacle refraction.

#### C. Initial ADD Selection

Note: A careful near-point ADD determination should be conducted prior to selecting a DAILIES TOTAL1® Multifocal (delefilcon A) trial lens.

The DAILIES TOTAL1® Multifocal (delefilcon A) lenses 3 ADD SYSTEM allows personalized fitting for presbyopic patients. The table below makes initial ADD selection easy.

#### **DAILIES TOTAL1® Multifocal Lenses ADD SELECTION**

| SPECTACLE ADD | BOTH EYES |
|----------------|-----------|
| Up to +1.25 | LO |
| +1.50 to +2.00 | MED |
| +2.25 to +2.50 | HI |

| Example 1: | OD | | os |
|-------------------------------------|------------------|--------|----------|
| Spherical Rx: | -4.50 -0.75 x 90 | | -4.00D |
| Spherical equivalent (least minus); | -4.75D | | -4.00D |
| Vertex corrected power: | -4.50D | | -4.00D |
| Spectacle Add: | | +0.75D | |
| Eye Dominance: | | OD | |
| Initial Trial Lens: | -4.50 LO | | -4.00 LO |
| CTD (4 = 0 0 0 | | | |

Example 2: OD os Spherical Rx: +4.25 -0.25 x 180 +4.00 D -0.50 x 180 Spherical equivalent +4.25D +3.75D (least minus): Vertex corrected +4.50D +3.75D power: Spectacle Add: +2.00D **Eye Dominance:** OS **Initial Trial Lens:** +4.50 MED +3.75 MED

#### 4. Initial Lens Fitting Evaluation

- a) Insert the lenses selected in Section 3 (above). If the exact power is not available, choose the next closest least minus/most plus lens power in your trial set.
- b) Allow the lenses to settle on the eyes for approximately 10 minutes. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate with the patient's tears.
- c) Evaluate the fit of the lenses on the eye. The **Push-up Test** as described below is an important part of the lens evaluation. The following guidelines will be helpful in evaluating the physical fit of the lens:

#### **Characteristics of a Well-fitted Lens**

A well-fitted DAILIES TOTAL1® Multifocal (delefilcon A) contact lens satisfies the following criteria:

- Full corneal coverage and good centration (no limbal exposure).
   A lens that is decentered > 1 mm, particularly temporal, is less likely to give adequate vision.
- Lens movement of 0.1 to 0.5 mm should be present to allow tear exchange under the lens during a blink in primary gaze or upward gaze and to avoid variable vision.

#### Push-up Test:

- This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then pull the lid back down and observe the return of the lens.
- A well fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- 3. Good comfort.
- 4. Acceptable visual acuity with over-refraction.

#### Characteristics of a Tight (Steep) Lens Fit

A tight or steep fit should not be dispensed. If a lens fit is judged to be too steep a flatter lens (larger base curve), if available, should be evaluated. A tight or steep lens fit would display some or all of the following characteristics:

- 1. Good centration.
- Insufficient or no lens movement during a blink in primary gaze or upward gaze.
- Excessive conjunctival drag (visible movement of the conjunctival vessels when the lens moves during a blink or during the push-up test). Note: presbyopes often have loose conjunctiva, some conjunctival movement is occasionally seen and may not be a sign of a tight fit. See Push-up Test below.

#### Push-up Test:

- A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- 4. Good comfort.
- 5. Blurred vision between blinks.

#### Characteristics of a Loose (Flat) Lens Fit

If a lens fit is judged to be too flat a steeper lens (smaller base curve), if available, should be evaluated. A loose lens fit would display some or all of the following characteristics:

- 1. Decentration.
- Excessive lens movement during the blink in primary or upward gaze.

#### Push-up Test:

- A loose fitting lens will move very easily, well beyond the limbus and possibly encroaching upon or going beyond the pupil. It will then return very quickly to its original position and often times return lower than its original position.
- 3. Reduced comfort.
- 4. Lens edge standoff.
- 5. Blurred vision immediately after the blink.

#### 5. Initial Lens Visual Evaluation

While lenses are settling, it is helpful to take the patient from the exam room to a "real-world" setting such as a room with an outside view. Once an acceptable fit has been achieved, the visual performance of the lenses may be evaluated. Visual acuity is tested at distance. If necessary, a spherical over-refraction should be performed using a trial frame or hand held lenses rather than a phoropter. This technique is essential when fitting multifocal lenses because it allows the patient to maintain the head posture and direction of gaze (relationship between eye and head) that he or she would naturally use during everyday tasks. This ensures that the visual performance of the lens is being assessed under conditions where the on-eye positioning matches that which will occur when the lens is being used, for example, for near work activities. In addition, pupil size will not be artificially increased

by the reduction in light associated with looking through the aperture of the phoropter cells, or decreased by proximal cues associated with the nearness of the instrument.

#### 6. Fitting Procedures

<u>Step 1</u>: After the trial lenses have settled for approximately 10 minutes, measure distance acuity while the patient is viewing the chart binocularly (i.e., simultaneously with both eyes). Next, evaluate the patient's subjective impression of the near vision when trying to read typical everyday material (e.g., a newspaper, magazine, and cell phone). Lighting and reading distance should be what is normal for the patient.

<u>Step 2</u>: If distance or near vision is unsatisfactory, perform a *binocular distance* over-refraction, as follows. Use hand-held trial lenses and encourage plus. For example, if a Plano and +0.25D over-refraction yields the same results, use the +0.25D endpoint. Re-check visual acuity and visual quality as described in Step 1 above. If over-refraction is other than plano, go immediately to new trial lenses, keeping ADD the same.

Step 3: If distance and near vision are satisfactory, dispense lenses and remind patient to use good light when reading fine print or use additional reading glasses if needed. It is helpful to let the patient experience the lenses in their natural environment before further procedures for enhancing vision are performed.

<u>Step 4</u>: **Enhanced Near Vision.** If near vision is unsatisfactory, determine the dominant eye by the following method. Determine the eye with **greatest plus acceptance** by placing +1.50 handheld trial lens over each eye alternately while patient views in the distance with both eyes open. Consider the eye for which binocular vision blurs *least* with the +1.50 to be the non-dominant eye. Other methods to determine the dominant eye are appropriate.

<u>Step 4A:</u> Check the patient's binocular acuity with +0.50 over the non-dominant eye to determine if near vision is improved and distance vision is still acceptable. If so, place a new trial lens with the same ADD on the non-dominant eye, adjusting the distance power by +0.50.

| Enhanced near vision, Step A | | |
|---|---|---|
| SPECTACLE ADD | SPECTACLE ADD DOMINANT EYE | |
| Up to +1.25 | LO | with additional +0.50 |
| +1.50 to +2.00 | MED | with additional +0.50 |
| +2.25 to +2.50 | HI | with additional +0.50 |

Next, re-check visual acuity and visual quality as described in Step 1 above. If satisfactory, dispense new distance lens power for the non-dominant eye. If near vision is still unsatisfactory, proceed to Step B:

Step 4B: If near vision is still unsatisfactory, adjust ADD as shown below.

| Enhanced near vision, Step B | | |
|---|---|---|
| SPECTACLE ADD | NON-DOMINANT EYE<br>(PLUS ACCEPTED) | |
| Up to +1.25 | MED | MED |
| +1.50 to +2.00 | MED | HI |
| +2.25 to +2.50 | HI | MED |

Note: It is common to question the rather non-intuitive step we suggest for enhancing vision at near in the HI ADD range, where the suggestion is to "back off" to a MED ADD for the non-dominant eye, the same suggestion we make for enhancing distance vision (below). The reason for this is that after establishing (in Step A) that increasing plus is not helpful, the next most common reason for blur at near (or distance) is unacceptable ghosting that degrades the image quality. Backing down to the MED ADD in one eye can often relieve that and actually improve vision at near.

<u>Step 5</u>: Enhanced Distance Vision. If distance over-refraction did not improve visual acuity, adjust ADD according to the chart below.

| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE<br>(PLUS ACCEPTED) |
|----------------|--------------|-------------------------------------|
| +1.50 to +2.00 | Lo | MED |
| +2.25 to +2.50 | HI | MED |

#### FITTING GUIDELINES (Monovision)

#### **Patient Selection**

#### A. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. Patients with reduced visual acuity, such as the amblyopic patient, may not be a good candidate for monovision.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it must be determined by trial whether this patient can function adequately with monovision. Monovision contact lens wear may not be optimal for such activities as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- driving automobiles (e.g., driving at night). Patients who cannot
  pass requirements for a driver's license with monovision
  correction should not drive with this correction. An additional
  over-correction can be prescribed to improve vision.

#### B. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with bifocal reading glasses. Each patient must understand that monovision, as well as other presbyopic contact lenses, or other alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision in straight-ahead and upward gaze that monovision contact lenses provide compared to spectacle bifocals.

#### **Eye Selection**

Generally, the non-dominant eye is corrected for near vision. The following test for eye dominance can be used:

#### A). Ocular Preference Determination Methods

- Method 1 Determine which eye is the "sight eye". Have the
  patient point to an object at the far end of the room. Cover
  one eye. If the patient is still pointing directly at the object,
  the eye being used is the dominant (sighting) eye.
- Method 2 Determine which eye will accept the added power for near with the least reduction in distance vision. Place a trial spectacle near ADD lens in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

#### B). Refractive Error Method

 For anisometropic corrections, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

#### C). Visual Demands Method

 Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

#### Example:

A person who places copy to the left side of the desk will usually function best with the near lens on the left eye.

#### **Special Fitting Considerations**

#### **Unilateral Lens Correction**

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens while a bilateral myope may require only a distance lens.

- Examples:
- **Emmetrope:** A presbyopic emmetropic patient who requires a +1.75 diopter ADD would have a +1.75 lens on the near eye and the other eye left without a lens.
- Bilateral myope: A presbyopic patient requiring a +1.50 diopter ADD who is -2.50 diopters myopic in the right eye and -1.50 diopters myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.
- Unilateral astigmat:
  - a) Emmetropic in one eye, astigmatic in the other

| Spectacle Rx | Potential Monovision Rx |
|---------------------|----------------------------|
| O.D. Plano | Uncorrected for distance |
| O.S1.00 -1.00 x 090 | +0.50 -1.00 x 090 for near |
| Add: +1.50 | |

b) Myopic in one eye, astigmatic in the other

| Spectacle RX | Potential Monovision RX |
|---------------------|--------------------------------|
| O.D1.50 | Uncorrected for near |
| O.S2.00 -1.75 x 090 | -2.00 -1.75 x 090 for distance |

#### **Amblyopia**

The amblyopic patient may not be a good candidate for monovision. **Astigmatism** 

Patients with less than 1.50 diopters of astigmatism might be successfully fit in DAILIES TOTAL1® (delefilcon A) spherical lenses.

- Determine which eye to use for the near prescription (see Eye Selection, A-C. above)
- Add the appropriate near add power to the spherical component of the astigmatic prescription for that eye.


Example: Spectacle Rx Potential Monovision Rx

O.D.: -2.50 -0.75 x 180 -2.50 -0.75 x 180 for distance

O.S.: -3.00 -1.75 x 165 -2.00 -1.75 x 165 for near

Add: +1.00

Dominant eye: O.D.

#### **Near Add Determination**

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

#### **Trial Lens Fitting**

A trial lens fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the directions in the *General Fitting Guidelines and Base Curve Selection* described earlier in the guide.

Case history and standard clinical evaluation procedures should be used to determine the suitability of monovision. Determine which eye is to be corrected for distance and which eye is to be corrected for near. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Immediately after the correct power lenses are in place, walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tasks are completed, should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to news print and finally smaller type sizes.

After evaluating the patient's performance under the above conditions, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a less favorable prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

#### Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a few minutes or for several weeks. The longer these symptoms persist, the poorer the chance for successful adaptation. To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it is recommended that patients be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several

weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive under optimal driving conditions. After adaptation, and success with these activities, the patient should be able to drive under other conditions with caution.

#### **Other Suggestions**

The success of the monovision technique may be further improved by having your patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Have supplemental spectacles to wear over the monovision contact lenses for specific visual tasks. This is particularly applicable for those patients who cannot meet driver's licensing requirements with a monovision correction.
- Make use of proper illumination when carrying out visual tasks.

Success in fitting monovision can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of the clear near vision in straight ahead and upward gaze with monovision.

The decision to fit a patient with a monovision correction is most appropriately left to the eye care professional in conjunction with the patient after carefully considering the patient's needs. All patients should be supplied with a copy of the **Patient Instruction Booklet**, which contains important instructions for the monovision wearer. You can obtain copies of the instruction book by calling customer service in the USA at (800) 241-5999.

#### **DISPENSING VISIT**

To help ensure patient success the following steps should be conducted with each patient, even if they have previously worn contact lenses. Even experienced wearers are prone to develop bad habits over time.

DAILIES TOTAL1® brand (delefilcon A) lenses are supplied sterile in foil sealed blister pack containers. Open the foil pack by peeling back the foil lidding material and gently slide the lens out of the container with your finger, or pour the lens onto the palm of your clean hand.

Conduct the following steps with each patient, even if they have previously worn contact lenses:

#### A. Verification of Lens Fit

Evaluate lens fit and visual response with the lens on the eye. The criteria of a well-fitted lens should be met and the patient's visual acuity should be acceptable. If not, the patient should be refitted with a more appropriate lens.

#### B. Hygiene and Lens Handling Instructions

Good hygiene and proper lens handling are important factors in achieving safe, comfortable lens wear. Instruct the patient on hygiene and handling of lenses. Patients who are unable to place and remove lenses should not be provided with them.

#### C. Lens Wear and Replacement Schedules (see Package Insert)

Prescribe and explain the daily disposable wear schedule. Explain that lenses are to be discarded after each daily wearing period. Determine the maximum suggested daily wearing period based on the patient's physiological eye condition. There may be a tendency for the patient to over-wear their lenses initially. For some patients who have never worn contact lenses consider a wearing schedule that allows for a gradual increase in wearing time.

#### D. Lens Care Directions (see Package Insert)

The lenses are not intended to be cleaned or disinfected and should be discarded after a single use. The eye care professional may recommend lens rewetting drops, as needed.

#### E. Specific Instructions for Presbyopic Patients

Specific instructions, explanations and demonstrations are important for optimizing patient success with multifocal contact lenses. The following information and instructions have proven useful in advising patients who wear DAILIES TOTAL1® Multifocal (delefilcon A) soft contact lenses.

- A contact lens that contains different powers for distance and near involves greater technological and optical complexity than does a bifocal or multifocal spectacle lens. This is because the contact lens moves with the eye, rather than having the eye move up and down while the lens remains suspended in a frame. While the contact lens therefore gives an unobstructed field of view and greater freedom regarding where to look, these advantages may mean that the sharpness of vision may not always be exactly the same as what would be experienced with spectacles.
- Although many individuals use DAILIES TOTAL1® Multifocal (delefilcon A) contact lenses for full-time wear, it is not unusual to find that there may be some activities where one prefers to CR-6479, v 3.0

wear spectacles, or where the disadvantages associated with spectacles are outweighed by other issues. This is an entirely normal and natural response to the challenges presented by presbyopia.

- Situations where vision with multifocal contact lenses may be less sharp or otherwise "different" than what is experienced with spectacles often involve low illumination (e.g., a semi-dark room), reduced visibility (e.g., outdoor conditions of fog or heavy rain), or isolated sources of very bright light (e.g., headlights of an oncoming vehicle on a narrow country road). Patients should be instructed to make use of good light when reading fine print.
- Patients should be aware that it might be advisable to refrain from wearing their lenses while driving, flying an airplane or operating heavy machinery while wearing their lenses until they gain some experience with the lenses in a similar visual environment.
- Small changes in lens power can often make a significant difference in the quality of the vision experienced with multifocal contact lenses. Such changes can be best tailored to individual needs and environmental conditions that the patient will personally encounter on a day-to-day basis. Confidence and assurance that such refinements, if needed, can be achieved are important for patient motivation during the initial period of lens wear.

#### F. Additional Instructions

Review the Package Insert

Provide the patient with all relevant information and precautions on the proper use of the lenses that are prescribed.

 Provide the Patient Instruction Booklet for DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) Contact Lenses.

Give the patient a copy of the *Patient Instruction Booklet* for DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) soft contact lenses. Review the contents so the patient clearly understands the prescribed lens wear, care, and replacement schedule. In the USA you can obtain copies of the instruction book by calling Alcon customer service at (800) 241-5999.

#### **Follow-Up Examinations**

Follow-up care is extremely important for continued successful contact lens wear. Follow-up care should include:

- Case history, including questions to identify any problems related to contact lens wear
- Management of specific problems, if any, and
- A review with the patient of the lens wearing schedule, replacement schedule and handling procedures.

#### Follow-up Examination Procedures

Patients should be instructed to wear lenses prior to a follow-up examination.

CR-6479, v 3.0




- Record patient's symptoms, if any.
- Measure visual acuity monocularly and binocularly with the contact lenses in place.
- · Perform an over-refraction to check for residual refractive error.
- · With a biomicroscope, evaluate lens fitting.
- Remove the lenses and conduct a thorough biomicroscopic examination with fluorescein. Rinse eyes with saline before re-inserting lenses.
- Evert upper lids to determine condition of tarsal conjunctiva.
- Periodically perform keratometry and spectacle refractions. These results should be recorded to compare to the initial measurements.
- If any observations are abnormal, use professional judgment to manage the problem and restore the eye to optimal conditions. If visual requirements are not satisfied during any follow-up examination, the patient should be re-fitted with a more appropriate lens.

#### **LENS HANDLING HINTS**

#### **Lens Insertion**

- When about to place the lens on the eye, make sure the lens sits up on the placement finger. The finger should be dry so surface tension does not cause the lens to adhere to the finger.
- Check to see that the lens is right side out. A lens that is placed on the eye inside out may not feel comfortable or provide good vision.

One way to do this is to perform the 'taco test' by placing the lens between your thumb and index finger and squeeze the edges together gently.

- If the edges come together, the lens is right side out.
- If the edges turn outward, the lens is wrong side out. Carefully reverse it with your fingers.



Another way is to place the lens on the tip of your index finger and check its shape.

- If the edge appears bowl-shaped, it is right side out.
- If the edge has a lip or flares outward, it is wrong side out and must be reversed.
- Place the lens directly onto the cornea (placing it on the lower sclera can lead to the lens folding after a blink). While continuing to hold both lids in place, the patient should look down to seat the lens. The lids may then be released.




#### Lens Removal

- Wash hands thoroughly with soap that does not have any oils, lotions or perfumes.
- Carefully dry hands with a lint-free towel.

It is important to remind patients to **dry their hands thoroughly** prior to removing their lenses. The surface of DAILIES TOTAL1® brand lenses is designed to stay very wet and lubricious, or slippery while on the eye. If their fingertips are wet they are likely to slip across the surface of the lens making removal more difficult.

- Slide the lens off the cornea (down or to the side) onto the sclera. This
  produces a fold in the lens, which assists in removal. With the index finger
  and thumb, gently pinch the lens off the eye.
- Discard lenses.

#### Care for a Sticking Lens

In the unlikely event that the lens sticks (stops moving) or begins to dry
on the eye, instruct the patient to apply several drops of a recommended
lubricating solution (used in accordance with package labeling). The
patient should wait until the lens begins to move freely on the eye before
attempting to remove it. If the lens continues to stick, the patient should
immediately consult the eye care professional.

#### IN OFFICE CARE OF TRIAL LENSES

Eye care professionals should understand and educate contact lens technicians concerning proper use of trial lenses.

- Each contact lens is shipped sterile in a sealed blister pack containing phosphate buffered saline with additives. Hands should be thoroughly washed and rinsed and dried with a lint-free towel prior to handling a lens. In order to insure sterility, the blister pack should not be opened until immediately prior to use.
- Delefilcon A lenses are for daily disposable wear only and should be discarded after a single use. The lenses should be disposed of after a single use and not be re-used from patient to patient.

#### **DISPOSAL AND RECYCLING**

Dispose of contact lenses and the blister pack lidding in the waste bin, not down the sink or toilet. The carton packaging and the polypropylene (PP) plastic shell of the blister pack should be placed in the waste bin or recycled according to local waste management guidance.

#### ADDITIONAL INFORMATION

For assistance with fitting or clinical questions regarding DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal contact lenses eye care professionals having questions or problems should contact Medical Information Systems in the USA at (800) 241-7468. To order DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal contact lenses contact your Alcon sales representative or call Customer Service, in the USA at (800) 241-5999.

CR-6479, v 3.0


#### Alcon

#### DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) soft contact lenses for Daily Disposable Wear

900236420

important. This package insert is effective as of December 2019 and applicable to the deletflicon A contact lenses described below. Please read carefully and keep this information for future up ordessional, but should be made available to patients upon request. The eye care professional should provide the patient with appropriate instructions that pretain to the patient's prescribed a decayer from Actor by examing Constructions and a 1-80-024-1-9990 ordinated from a very section of adultion. a Patient Instruction Dockeler's available in servementaries of a work and ordination and a very service and ordination and d for the eye care



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional.

#### PRODUCT DESCRIPTION

DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilcon A) soft contact lenses are made from a lens material that is 33% Ny sort contact relates are intact or maken a material material water and 67% (delefficen A) polymer, a silicone containing hydrogel with added phosphatidylcholine. The core lens material containing 33% water transitions through a water gradient to a hydrogel surface layer that exceeds 80% water. Lenses contain the color additive copper phthalocyanine, a light blue tint, which makes them easier to see when handling.

#### Lens Properties

Refractive Index hydrated: 1.42

93% (@ 610 nm, -1.00 D) 140 x 10<sup>-11</sup> (cm²/sec)(ml 0<sub>2</sub> /ml x mm Hg), measured at 35° C Light Transmittance:
 Oxygen Permeability (Dk):

(intrinsic Dk-Coulometric method)

· Water Content: 33% by weight in normal saline

#### Surface Water Content:

Lens Parameters • Diameter Range 13.0 to 15.0 mm
• Spherical Power Range -20.00 to +20.00 D
• Base Curve Range 8.0 to 9.2 mm

#### DAILIES TOTAL1® (delefilcon A) spherical contact lenses

Chord Diameter:
 Center Thickness:

0.09 mm @ -3.00 D (varies with power) 8.5 mm Rase Curve:

-0.50 to -6.00 D (0.25 D steps) -6.50 to -12.00 D (0.50 D steps) +0.50 to +6.00 D (0.25 D stens)

#### DAILIES TOTAL1® Multifocal (delefilcon A) contact lenses

14.1 mm 0.09 mm @ -3.00 D (varies with Chord Diameter:
 Center Thickness:

 Base Curve:
 Powers: 8.5 mm +6.00 D to -10.00 D (0.25 D steps) ADD: LO. MED. HI

NOTE: Hereafter, DAILIES TOTAL1® spherical contact lenses and DAILIES TOTAL1® Multifocal contact lenses will simply be referred to as delefilcon A contact lenses unless product distinction is necessary.

#### ACTIONS

When hydrated and placed on the comea, **delefilcon A** contact lenses act as a refracting medium to focus light rays on the

#### INDICATIONS (Uses)

DAILIES TOTAL1® (delefilcon A) spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

DAILIES TOTAL1® Multifocal (delefilcon A) soft contact lenses Database Total: Immittoda (uderticon y source) are indicated for the optical correction of refractive ametropia (myopia and hyperopia) and/or presbyopia in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 (D) or less and who may have up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

The lenses are to be prescribed for single use, daily disposable wear. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

#### CONTRAINDICATIONS (Reasons Not To Use) DO NOT use delefilcon A contact lenses when any of the following exists:

 Inflammation or infection of the anterior chamber of the eye
 Active disease, injury or abnormality affecting the cornea, conjunctiva, or evelids

CR-6479, v 3.0

- Microbial infection of the eye
   Insufficiency of lacrimal secretion (dry eye) that interferes with contact lens wear
   Corneal hypoesthesia (reduced corneal sensitivity)
- Use of any medication that is contraindicated or interferes
- with contact lens wear, including eve medications Any systemic disease which may be exacerbated by or
- interferes with contact lens wear Allergic reactions or ocular irritation of the ocular surfaces or adnexa that may be caused by or exaggerated by the wearing of contact lenses
- Detaint history of recurring eye or eyelid infections, adverse effects associated with contact lens wear, intolerance or abnormal ocular response to contact lens wear
- · If eves become red or irritated

#### WARNINGS

#### Advise patients of the following warnings pertaining to

- contact lens wear:

  Problems with contact lenses and lens care products could result in serious injury to the eye. It is essential that patients follow their eye care professional's directions and all labeling instructions for proper use of lenses and lens care products.

  Serious eye problems, including corneal ulcers, can
- develop rapidly and lead to loss of vision.

  Daily wear lenses are not indicated for overnight wear, and patients should be instructed not to wear lenses while sleeping. Clinical study results have shown that the risk of serious adverse reactions is increased when contact lenses
- Studies² have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than ionsmokers.
- If a patient experiences eve discomfort, foreign body in a patient experiences eye discounting, relegiously sensation, excessive tearing, vision changes, or redness of the eye, the patient should be instructed to immediately remove lenses and promptly contact his or her eye care professional. It is recommended that contact lens wearers see their eve care professional regularly as directed.

To prevent damage to the eyes or to the contact lenses, the following precautions should be taken:

Special Precautions for the Eye Care Professional Due to the small number of patients enrolled in the clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the eye care professional should consider all characteristics of the lens

that can affect lens performance and ocular health, including oxygen permeability, central and peripheral thickness and optic zone diameter. The potential impact of these factors on the patient's ocular he potential implact or unless factors on the patients scelar health should be carefully weighed against the patient's need for refractive correction; therefore the continuing ocular health of the patient and lens performance on the eye should be carefully evaluated on initial dispensing and monitored on an ongoing

- basis by the prescribing eve care professional. Fluorescein, a yellow dye, should not be used while the lenses are on the patient's eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used, the eyes should be flushed thoroughly with sterile saline solution that is recommended for in eve use prior to inserting lenses. Avoid dispension saline from an aerosol can directly into the eve
- Patients who wear contact lenses to correct presbyopia may not achieve the best possible corrected visual acuity for eithe far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient
- Before leaving the eye care professional's office, the patient should be able to promptly remove their lenses or should have someone else available who can remove their lenses for them.
  Eve care professionals should instruct the patient to remove
- the lenses immediately if the eye becomes red or irritated
- · Routine eye examinations are necessary to help assure the continued health of the patient's eyes. Eye care professionals should make arrangements with the patient for appropriate follow-up visits. Alcon recommends that patients see their e care professional once each year, or more often, as recommended by the eye care professional.

- . Diabetics may have reduced corneal sensitivity and thus are more prone to corneal injury and do not heal as quickly or ompletely as non-diabetics.
  isual changes or changes in lens tolerance may occur during
- pregnancy or use of oral contraceptives. Caution patients

#### Eye Care Professionals should carefully instruct patients about the following safety precautions:

#### Handling Precautions

Be sure that before leaving the eye care professional's office
 the patient is able to promptly remove lenses or have
 someone else available to remove them.

- . Good hygiene habits help promote safe and comfortable lens wear. Always wash, rinse and thoroughly dry hands with a lint-free towel before handling lenses.

  REMOVE A LENS IMMEDIATELY if an eye becomes red or
- irritated.
- · Always handle lenses carefully. Never use tweezers or other sharp objects such as fingernalis to remove lenses from the lens container unless specifically indicated for that use. Do not use if blister package is damaged or not sealed
- completely. This may result in product contamination which can lead to a serious eve infection
- Ensure that the correct lens for each eye is available. Shake the blister pack gently prior to opening. Remove the lens from the blister pack by carefully pouring the lens onto the palm of your clean hand. Ensure the lens is right side out. Inspect enses prior to insertion. Do not insert damaged lenses
- To insert lenses:

   Wash and rinse hands thoroughly and dry completely with a clean, lint free towel before handling lenses.
- Place a lens on the tip of your clean and dry right or left index finger, place the middle finger of the same hand close to lower eyelashes and pull down the lower eyelid. Use the fingers of the other hand to lift the upper eyelid.
- Place the lens directly on the eye (cornea) and gently roll
- finger away from the lens Look down and slowly remove the hand, releasing the lower
- Look straight ahead and slowly remove the other hand,
- releasing the upper lid. Blink gently.
- To remove lenses:
   Wash and rinse hands thoroughly and dry completely with a clean, lint free towel before handling lenses. Make sure hands are clean and completely dry.
- Rlink fully several times
- While looking up, slide the lens down onto the white part of the eye.
- Remove the lens by pinching gently between the thumb and
- forefinger. Do not pinch the eye tissue.

  If the lens is difficult to grasp, dry fingers once more and try again. Do not use rewetting drops in this instance.
- f a lens decenters on the eye, it may be possible to recenter it by:

- Closing the eye and massaging the lens into place, or Looking in the direction of the lens and blinking gently, or Gently pushing the off-centered lens onto the cornea with light finger pressure on the edge of the upper or lower
- If a lens tears in the eye it will feel uncomfortable. Advise wearers it is impossible to lose a contact lens or part of a contact lens behind the eye and to remain calm. Lens pieces may be removed by pinching them as for normal lens removal, carefully avoiding pinching the eye tissue. If the lens pieces do not seem to remove easily, rinsing with saline is recommended. If this does not help, the wearer should contact an eye care professional for assistance

#### Lens Wearing Precautions:

- Patients should never exceed the prescribed wearing schedule regardless of how comfortable the lenses feel. Doing so may increase the risk of adverse effects.
- The lens should move freely on the eve at all times. If the lens sticks (stops moving) on the eye, follow the recommended directions in the Care for a Sticking Lens section. If non-movement of the lens continues, the patient should be
- instructed to consult their eye care professional immediately. The eye care professional should be consulted about wearing lenses during water sports and water related activities.

  Exposure to water or other non-sterile liquids while wearing


- contact lenses in activities such as swimming, water skiing, and hot tubs may increase the risk of ocular infection, including but not limited to Acantamacela keratitis. Never allow contact lenses to come into contact with non-sterile liquids (including have whater and salive) as microbi contamination can occur, which may lead to permanent eye
- eye irritation, infection, or lens damage may result if
- cosmetics, lotion, soap, cream, hair spray, deodorant, aerosol products or foreign particles come in contact with lenses.

  Environmental fumes, smoke, and vapors should be avoided in order to reduce the chance of lens contamination or physical
- trauma to the cornea.

   Lenses should be disposed of each day upon removal from the
- eye.
  Discard any lens which has become dehydrated or damaged.
- Replace with a sterile, fresh, new lens.

  Note the correct lens power for each eye to prevent getting
- them mixed up.

  Always carry spare lenses with you or have back-up spectacles available.
- Do not share lenses with anyone as this may spread micro-organisms which could result in serious eye health
- problems.
   Do not use lenses beyond their expiration date.

- Other Topics to Discuss with Patients:

   Periodic eye examinations are extremely important for contact lens werens. Schedule and conduct appropriate follow-up examinations to determine ocular response. Alcon recommends that patients see their eye care professional once each year or as recommended by the eye care professional.
- professional.

  Certain medications may cause dryness of the eye, increased lens awareness, lens intolerance, and blurred vision or visual changes. These include, but are not limited to, antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sckness. Caution patients using outher medications accordingly and prescribe proper remedial
- Presented the contract of the accordingly.

# Who Should Know that the Patient is Wearing Contact Lenses:

- Lenses:

  Patients should inform their health care practitioners that they are wearing contact lenses.

  Patients should inform their employers that they are wearing contact lenses. Some jobs may require the use of eye protection equipment or may require that contact lenses not be worn.

It is strongly recommended that patients be provided with a co of the DAILIES TOTAL1® and DAILIES TOTAL1® Multifocal (delefilion A) Contact Lenses Patient Instruction Booklet availal from Alcon and understand its contents prior to dispensing the

#### WATER ACTIVITIES

Do not expose contact lenses to water while wearing them.

Utility explose curricus views that can lead to severe infection, vision loss or blindness. If lenses have been submersed in water when showering or swimming, discard them and replace with a new pair, Ask the Eye Care Professional for recommendations about wearing lenses during any activity

ADVERSE EFFECTS
Patients should be instructed to check eyes regularly to make sure they look well, feel comfortable and vision is clear. Potentially serious complications are usually clear. Potentially serious complications are usually accompanied by one or more of the following signs or symptoms:

• Moderate to severe eye pain not relieved by removing the lens Foreign body sensation

• Excessive watering or other eye secretions including mucopurulent discharge

• Redness of the eyes

• Photophobia (light sensitivity)

• Burning, stinging or tiching or other pain associated with the eyes

- Comfort is less compared to when the lens was first placed on
- eye Poor visual acuity (reduced sharpness of vision)
- Blurred vision, rainbows or halos around objects
   Feeling of dryness

#### WHAT TO DO IF A PROBLEM OCCURS Patients should be instructed that if any of the above signs

#### or symptoms are noticed, he or she should: • IMMEDIATELY REMOVE THE LENSES.

- IMMEDIATELY REMOVE THE LENSES.
  If the disconfort or problem stops, discard the lens and replace it with a new one.
  If the disconfort or problem continues after removing lens(es) or upon insertion of a new lens, IMMEDIATELY remove the lens(es) and contact the eye care professiona for identification of the problem and prompt treatment to
- for identification of the prouven any proups avoid serious yes demage.

  The patient should be informed that a serious condition such as comeal uden, interestion, comeal vascuslarization, or intis may be present, and may progress rapidly, Less serious reactions such as abarsaions, infillitates, and bacterial conjunctivitis must be managed and treated acrefully to avoid more serious complications.

  Additionally, contact lens wear may be associated with outlar these their rangine consideration of discontinuation or
- Additionally, Contact sens wear may be associated with occurs changes that require consideration of discontinuation or restriction of wear. These include but are not limited to local or generalized corneal edema, epithelial microcysts, epithelial staining, infiltrates, neovascularization, endothelial generalized corneal edema, epithelial microcysts, epithelial staining, infiltrates, neovascularization, endothelial polymegathism, tarsal papillary changes, conjunctival injection

#### ADVERSE EFFECT REPORTING

If a patient experiences any serious adverse effects associated with the use of DALLES TOTAL 1º brand (delefilicon A) contact lenses, please notify: Alcon Medical Safety in the USA at 1-800-757-9780.

#### FITTING GUIDE AND PATIENT BOOKLET

TITING GUIDE AND PATIENT BOOKLET

Onventional methods of fitting contact lenses apply to deleficon

tontact lenses. For a detailed description of the fitting

chiques, refer to the DAILES TOTAL1\*

Symbol/Abbreviation Description techniques, refer to the DAILIES TOTAL1\* and DAILIES TOTAL Multificaci (delelicon A) Contact Lenses Professional Fitting Information Guide. Both the professional fitting guide and a patient instruction booklet are available free of charge from: Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX, USA 76134-2099 1 and 241 English

#### LENS WEAR & REPLACEMENT SCHEDULES DAILY WEAR (less than 24 hours, while awak

- ALLY WEAR (less than 24 hours, while awake):

  To avoid tendency of the daily war patient to over-wear the lenses initially, stress the importance of adhering to a proper, initial wearing schedule. Normal daily wear of lenses assumes a minimum of 5 hours of non lers wear per 24 hour period. It may be advisible for patients who have never worn contact lenses previously to be given a wearing schedule that gradually increases wearing time over a few days. This allows more gradual advisable was wearing time over a few days. This allows more gradual advisable of the ocular tissues to contact lens wear.
- wear.

  The maximum daily wearing time should be determined by the eye care professional based upon the patient's physiological eye condition because individual responses to conduct losses vary. There may be a tendency for patients to over-wear the lenses initially. The eye care professional should stress the importance of adhering to the initial maximum wearing schedule. Studies have not been conducted to show that defellicon A contract lenses are also the war during sleep.
- deletion A contact tenses are safe to wear during sleep, therefore patients should be advised to remove their l'enses while sleeping. Normal daily wear of lenses assumes a minimum of 6 hours of non-lens wear per 24 hour period. Optimum individual wearing schedule will vary. Deletilion A contact lenses are intended to be worn once (daily disposable wear) and then discarded at the end of each wearing period. The patient should be instructed to start the next wearing period with a fresh new lens.

EMERGENCY LENS CARE
Cleaning and disinfection of daily disposable lenses is not recommended. The patient should be reminded to have replacement lenses or back-up spectacles available at all times.

CARE FOR A STICKING LENS
If the lens sticks (stops moving) or begins to dry on the eye,
instruct the patient to apply several drops of a recommended
lubricating solution (used in accordance with package labeling
fine patient should wait until the lens begins to more from
the eye before attempting to remove it. It is important that the
patient wash and dry their hands thoroughly before removing t
lens. If the lens continues to stick, the patient should IMMEDIATELY consult the eye care professional

# 

Eye care professionals should educate contact reas technicians concerning proper use of trial lenses. Each contact lens is shipped sterile in a blister pack containing phosphate buffered saline solution. Hands should be thoroughly washed and rinsed and dried with a lint-free towel prior to handling a lens. In order to ensure sterility, the blister pack

should not be opened until immediately prior to use. For fitting and diagnostic purposes lenses should be disposed of after a single use and not be re-used from patient to patient.

EMERGENCIES
The natient should be informed that if chemicals of any kind

Ehterman.
The galent should be informed used.
(nousehold products, gardening solutions, laboratory cnements)
etc.) are spiked into the eyes, the patient should.

Solution and immediately contact the eye care
professional or visit a hospital emergency room without

DISPOSAL AND RECYCLING
Dispose of contact lenses and the blister pack lidding in the Dispose of contact lenses and the blister pack number in unity of the waste bin, not down the sink or tollet. The carton packaging and the polypropylene (PP) plastic shell of the blister pack should be placed in the waste bin or recycled according to local waste management guidance.

#### HOW SUPPLIED

HOW SUPPLIED Each lens is packaged in a foil-sealed plastic container containing phosphate buffered saline solution with approximately 0.3% of polymeric wetting agents consisting of copolymes of polyamidoamine and polylacrylamide-acyfic) acid and is steam settilized. The package is marked with the base curve, diameter, dioptric power (and ADD power for multifacel lenses) manufacturing of number, date of manufacture, and expiration

| (B) only | CAUTION: Federal law (United States) restricts this device to sale by or on<br>the order of a licensed eye care professional. |
|---|---|
| 0 | Single sterile barrier system |
| STERILE | Sterilized using steam |
| | Use-by date (Expiry date) |
| LOT | Batch code |
| en | Two letter code for the language (Example shown: English) |
| (2) | Do not re-use |
| (9) | Do not use if blister package is damaged |
| DIA | Diameter |
| BC | Base curve |
| PWR | Power |
| L | Left |
| R | Right |
| D | Diopter (lens power) |
| ADD | Addition power |
| MAX ADD | Maximum effective addition power |
| L0 | Low |
| MED | Medium |
| HI | High |
| C€ | European conformity mark |
| Δ | Caution |
| (Ii) | Consult instructions for use |
| EO PEP | Authorized representative in the European Community |
| | Manufacturer |
| ₩ | Date of manufacture |
| MD Medical device | |
| 0 | Packaging waste license sign |

Manufacturer: Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX, USA 76134-2099

1-800-241-5999

www.alcon.com

U.S. Pat.: www.alconpatents.com

#### Alcon

© 2019 Alcon Inc.

Check for actual product availability as additional parameters may be introduced over time.

may be introduced over time. \$Schein, OD, Glynn RJ, Pogio EC, Seddon JM, Kenyon KR. The Relative Risk of Ulcarative Keratitis Among Users of Daily Wear and Extended Wear Soft Contact lenses. N Eng J Med. 1989; 321 (12):773-783.

#### **VERTEX DISTANCE CONVERSION CHART**

For minus lenses, read left to right; for plus lenses, read right to left. (12 mm Vertex Distance)

| - | + | - | + | - | + | - | + |
|------|------|-------|-------|-------|-------|-------|-------|
| 4.00 | 3.87 | 7.50 | 6.87 | 12.00 | 10.37 | 19.00 | 15.50 |
| 4.25 | 4.00 | 7.62 | 7.00 | 12.50 | 10.75 | 19.25 | 15.62 |
| 4.50 | 4.25 | 7.75 | 7.12 | 12.75 | 11.00 | 19.25 | 15.75 |
| 4.75 | 4.50 | 7.87 | 7.25 | 13.00 | 11.25 | 19.75 | 16.00 |
| 5.00 | 4.75 | 8.00 | 7.37 | 13.50 | 11.50 | 20.00 | 16.12 |
| 5.12 | 4.87 | 8.12 | 7.50 | 13.75 | 11.75 | 20.25 | 16.25 |
| 5.37 | 5.00 | 8.25 | 7.62 | 14.00 | 12.00 | 20.50 | 16.50 |
| 5.50 | 5.12 | 8.50 | 7.75 | 14.25 | 12.25 | 20.75 | 16.62 |
| 5.62 | 5.25 | 8.75 | 8.00 | 14.75 | 12.50 | 21.00 | 16.75 |
| 5.75 | 5.37 | 9.00 | 8.25 | 15.00 | 12.75 | 21.25 | 17.00 |
| 5.87 | 5.50 | 9.25 | 8.37 | 15.50 | 12.75 | 21.75 | 17.25 |
| 6.00 | 5.62 | 9.50 | 8.62 | 15.75 | 13.25 | 22.25 | 17.50 |
| 6.12 | 5.75 | 9.75 | 8.75 | 16.25 | 13.50 | 22.50 | 17.75 |
| 6.37 | 5.87 | 10.00 | 9.00 | 16.75 | 13.75 | 23.00 | 18.00 |
| 6.50 | 6.00 | 10.25 | 9.12 | 17.00 | 14.00 | 23.50 | 18.25 |
| 6.62 | 6.12 | 10.50 | 9.25 | 17.25 | 14.25 | 23.75 | 18.50 |
| 6.75 | 6.25 | 10.75 | 9.37 | 17.62 | 14.37 | 24.25 | 18.75 |
| 6.87 | 6.37 | 11.00 | 9.62 | 18.00 | 14.50 | 24.75 | 19.00 |
| 7.00 | 6.50 | 11.25 | 9.75 | 18.12 | 14.75 | 25.00 | 19.25 |
| 7.12 | 6.62 | 11.50 | 10.00 | 18.50 | 15.00 | 25.50 | 19.50 |
| 7.37 | 6.75 | 11.75 | 10.25 | 18.75 | 15.25 | 26.00 | 19.75 |

This page intentionally left blank

# Alcon

Manufacturer: Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX, USA 76134-2099

www.alcon.com

© 2019 Alcon Inc.

December 2019

W900236422-1219

CR-6479, v 3.0




# Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

#### APPENDIX H: BINOCULAR OVER REFRACTION



## Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

# DETERMINATION OF NEAR ADDITION NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE LENS FITTING CHARACTERISTICS SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIVE ERROR BIOMICROSCOPY SCALE DISTANCE AND NEAR SNELLEN VISUAL ACUITY EVALUATION DISTANCE LOGMAR VISUAL ACUITY MEASURMENT PROCEDURE PATIENT REPORTED OUTCOMES VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION

# Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

### **DETERMINATION OF NEAR ADDITION**

Title: Determination of Near Addition

**Document Type:** 

Document Number: Revision Number: 5

Title: Determination of Near Addition

Document Type:

Document Number: Revision Number: 5

CR-6479, v 3.0


Page 2.015

**Document Type:** 

Document Number: 5
**Document Type:** 

Document Number: Revision Number: 5

, NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE

Document Number: Revision Number: 9

#### LENS FITTING CHARACTERISTICS

**Document Type:** 

**Document Number: Revision Number: 6**  Title: Lens Fitting Characteristics

**Document Type:** 

Document Number: Revision Number: 6

CR-6479, v 3.0


Document Type:

Document Number: 6

Revision Number: 6

Document Number: Revision Number: 6

, SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS

**Document Type:** 

Document Number: 4

CR-6479, v 3.0


DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIVE ERROR

Document Number: 5

BIOMICROSCOPY SCALE

| Title: | Biomicroscopy Sc | ale |
|-------------------------|------------------|---------------------|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 10 |



| Title: | Biomicroscopy Scale | | |
|-------------------------|---------------------|-------------------------|----|
| <b>Document Type:</b> | | | |
| <b>Document Number:</b> | | <b>Revision Number:</b> | 10 |

| Title: | Biomicroscopy So | cale |
|-------------------------|------------------|---------------------|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 10 |



| Title: | Biomicroscopy So | cale |
|-------------------------|------------------|---------------------|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 10 |



| Title: | Biomicroscopy Scale | |
|-------------------------|---------------------|---------------------|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 10 |



#### DISTANCE AND NEAR SNELLEN VISUAL ACUITY EVALUATION

DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE

| Title: | Distance LogMAR Visual Acuity Measurement Procedure | |
|---|---|---|
| Document Type: | | |
| <b>Document Number:</b> | | Revision Number: 5 |

| Title: | Distance LogMAR Visual Acuity Measurement Procedure | |
|---|---|---|
| Document Type: | | |
| Document Number: | | Revision Number: 5 |



| Title: | Distance LogMAR Visual Acuity Measurement Procedure |
|---|---|
| <b>Document Type:</b> | |
| <b>Document Number:</b> | Revision Number: 5 |

#### PATIENT REPORTED OUTCOMES

| Title: Document Type: Document Number: | Patient Reported Outcomes | |
|---|---|---|
| | | Revision Number: 3 |

Page 1 of 1
# Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

# VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

# Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

APPENDIX J: GUIDELINES FOR COVID-19 RISK MITIGATION

| Title: | Guidelines for C | OVID-19 Risk Mitigation |
|-------------------------|------------------|-------------------------|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

#### 1.0 PURPOSE

The purpose of this document is to provide guidelines for the re-opening or initiation of clinical study sites participating in Johnson & Johnson Vision Care, Inc. (JJVCI) clinical studies during the COVID-19 pandemic.

#### 2.0 SCOPE

This document provides guidelines for Johnson & Johnson Vision Care (JJVCI) to address the potential risks from COVID-19 to study subjects, investigators, study site staff, and monitors at study sites. The guidance provided in this document is in effect from the date of approval through the date of retirement of this Work Instruction. At a minimum, this Work Instruction will be reviewed and updated on a quarterly basis, as appropriate.

NOTE: Re-opening of sites outside of the US will be evaluated on a country by country basis subject to local health authority guidance.

# 3.0 **DEFINITIONS**

American Academy of Optometry (AAO): The American Academy of Optometry is an organization of optometrists based in Orlando, Florida. Its goal is to maintain and enhance excellence in optometric practice, by both promoting research and the dissemination of knowledge. The AAO holds an annual meeting, publishes a monthly scientific journal, gives credentials to optometrists through the fellowship process and publishes position statements.

American Optometric Association (AOA): The American Optometric Association, founded in 1898, is the leading authority on quality care and an advocate for our nation's health, representing more than 44,000 Doctors of Optometry (O.D.), optometric professionals, and optometry students. Doctor of Optometry take a leading role in patient care with respect to eye and vision care, as well as general health and well-being. As primary health care providers, Doctor of Optometry have extensive, ongoing training to examine, diagnose, treat and manage ocular disorders, diseases and injuries and systemic diseases that manifest in the eye. The American Optometric Association is a federation of state, student, and armed forces optometric associations. Through these affiliations, the AOA serves members consisting of optometrists, students of optometry, paraoptometric assistants and technicians. The AOA and its affiliates work to provide the public with quality vision and eye care.

**Centers for Disease Control and Prevention (CDC):** The Centers for Disease Control and Prevention is a national public health institute in the United States. It is a United States federal agency, under the Department of Health and Human Services, and is headquartered in Atlanta, Georgia.

**COVID-19:** Current outbreak of respiratory disease caused by a novel coronavirus. The virus has been named "SARS-CoV-2" and the disease it causes has been named "Coronavirus Disease 2019" (COVID-19).

Clinical Study: Voluntary research studies conducted in people and designed to answer specific questions about the safety or effectiveness of drugs, vaccines, other therapies, or new ways of using existing treatments. May also be called clinical trials, studies, research, trials, or protocols.

Clinical Study Site: Location where a clinical study is conducted, such as a doctor's office, university, or laboratory. Clinical studies are conducted by Investigators who are individual(s) responsible for the conduct of the clinical study at a study site. If a study is conducted by a team of individuals, the Investigator is the responsible leader of the team and may be called the Principal Investigator.

Clinical Operations Manager (COM): The Johnson & Johnson Vision Care (JJVCI) individual responsible for the overall management of a clinical trial.

| Title: | Guidelines for Co | DVID-19 Risk Mitigation |
|-------------------------|-------------------|-------------------------|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

**Monitor:** An individual designated to oversee the progress of a clinical study and ensure that it is conducted, recorded, and reported in accordance with the protocol, Standard Operating Procedures (SOPs), Good Clinical Practice (GCP), and applicable regulatory requirements.

**Medical Safety Officer (MSO):** Physician who has primary accountability in their product portfolio for product health and safety, and who serves as an independent medical voice for patient safety.

**Safety Management Team (SMT):** A cross-functional, collaborative team responsible for review, assessment and evaluation of medical safety data arising from any source throughout the product life cycle.

#### 4.0 GUIDANCE FOR STUDY DOCUMENTS

In alignment with recent health authority guidance, JJVCI is providing recommendations for study-related management in the event of disruption to the conduct of the clinical study. This guidance does not supersede any local or government requirements or the clinical judgement of the investigator to protect the health, safety and well-being of participants and site staff. If, at any time, a participant's safety is considered to be at risk, study intervention will be discontinued, and study follow-up will be conducted as outlined in the protocol.

During the COVID-19 pandemic, the additional risks listed below need to be considered for study participants and study personnel:

#### 4.1 Additional Risks Related to the COVID-19 Pandemic:

- The possible transmission of the Coronavirus infection and consequent complications, beyond the risk of adverse events due to the investigational device and/or procedures.
- The risk may be higher in an optometric clinical study because of the close contact the subject will have with health care professionals during the procedures and assessments (since the investigator must make the measurements close to the subject's face) and, in addition the need for multiple follow-up visits/exams which may expose the subject to other patients and/or healthcare professionals who might be transmitting the virus, even if they do not have symptoms.
- Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions, which may lead to delays in scheduled follow-up visits.
- Subjects experiencing an adverse event related to contact lens wear may receive delayed treatment
  due to COVID-19 restrictions. In this event, all assessments that can be conducted virtually will be
  completed by the investigator to determine the best course of treatment for the subject, including
  an unscheduled visit, up to discontinuation from the study, as appropriate.

If a study subject is found to have contracted COVID-19 during participation in a study, he/she will be discontinued from the study and followed until COVID-19 Adverse Event (AE) resolution.

To help minimize the above potential risks, JJVCI recommend reviewing/complying with local, state, and governmental guidance for COVID-19 risks.

JJVCI will provide the following study specific documents with language pertaining to COVID-19 risks:

#### 4.1.1 Informed Consent:

Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed Consent document:

| Title: | Guidelines for COVID-19 Risk Mit | igation |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

#### STUDY ASSOCIATED RISKS RELATED TO COVID-19 (CORONAVIRUS) PANDEMIC

It is important to note that this study will be conducted, at least in part, during the COVID-19 pandemic. As such, additional risks associated with the infection with COVID-19 exist for you. This is particularly important for this study due, in part, to the closeness of the doctor during the study examinations.

The potential effects of the disease are not fully known, at this time, and may include long-term serious health consequences. In severe cases, this may result in hospitalization and/or death. Based on current knowledge from the Centers for Disease Control and Prevention (CDC), those at high-risk for severe illness from COVID-19 include older adults and people with underlying medical conditions.

During this study, all appropriate measures will be taken to minimize risks including the use of personal protective equipment such as masks and gloves, as well as proper sanitization. This is in conformance to guidance from the CDC, local health departments, and the state and county in which the study doctor's office is located. However, these measures may not completely eliminate the risks associated with contracting COVID-19.

If you are found to have contracted COVID-19 or feel ill with flu-like symptoms during participation in the study, you will not be permitted to continue in-office study follow-up visits, but you will receive instructions and your condition will be monitored by the doctor and/or study staff.

## 4.1.2 COVID-19 Risk Control Checklist (Attachment-B):

Will include COVID-19 risk control methods that are required by a site to conduct JJVCI clinical studies. The risk controls are consistent with CDC, AOA, AAO Guidance. The Principal Investigator will review/sign the study specific checklist prior to the Site Initiation Meeting.

# 4.1.3 Protocol Compliance Investigator(s) Signature Page:

Will include a statement indicating that the Principal Investigator (PI) agrees to conduct the study in compliance with all local, state, and governmental guidance's for COVID-19 risk mitigation.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

# 4.1.4 Study Site Initiation Training Slides:

Will include suggestions to help mitigate potential transmission of COVID-19. Suggestions may include maintaining social distancing in the clinical site by staggered scheduling of study patients, wearing proper PPEs, frequent disinfection, and installing shields on the slit lamp and other applicable equipment.

#### 5.0 GUIDANCE FOR REMOTE SUBJECT VISITS

Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions. Possible disruption of the study as a result of COVID-19 control measures may lead to delays in scheduled follow-up visits.

Subjects may be delayed in being seen for study follow up visit(s), for example due to COVID-19 control measures or due to the subject's concerns or fears about COVID-19 risk. When appropriate, the remote assessment will be conducted to the extent possible. Discussions with the subject during remote assessments may include:

Document Type:

Document Number:

Revision Number: 5

| Procedure | Details |
|---|---|
| Subject Reported Ocular<br>Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire regarding the test article when applicable and feasible. |
| Change of Medical History<br>(Adverse Events) and<br>Concomitant Medications /<br>Therapies Review | Record any adverse events or medical history changes from the previous study visit with the subject/parents. Review the subject's concomitant medications/therapies and record any changes from the previous study visit. |
| Wearing Time and Compliance | Record the average wearing time (including number of hours per day during weekdays and weekends, and number of days per week). Confirm compliance with the prescribed wear schedule. Record and discuss the lens wear compliance based on the subject's self-report. For example, the subjects will be asked the time of the day the subject typically puts on the study lenses in the morning and takes off in the evening, the number of days per week lenses were worn, and the number of consecutive days the subject didn't wear the study lenses, etc. |

The discussion with the subject will be documented in EDC under Tele-Visit and a minor protocol deviation will be noted. If during the telephone consultation, a subject states he/she wishes to discontinue participating in the study, instruct the subject to stop wearing the study lenses and schedule the subject to return to the clinic for a Final Evaluation at the at earliest possible time. Subjects should return all unused lenses to the clinic at the last visit.

Changes in study visit schedules, missed visits, or participant discontinuations may lead to missing data, including data related to protocol-specified procedures. Case report forms should capture specific information regarding the basis of missing data, including the relationship to the COVID-19 pandemic.

#### 6.0 STUDY CONDUCT DURING PANDEMIC

It is recognized that the Coronavirus Disease 2019 (COVID-19) pandemic may have an impact on the conduct of this clinical study due to, for example, self-isolation/quarantine by participants and study-site personnel; travel restrictions/limited access to public places, including Optometry Clinics; and changes in clinic procedures required to address the COVID-19 challenge.

Every effort should be made to adhere to protocol-specified assessments for study participants, including follow-up. However, if scheduled visits cannot be conducted in person at the study site it is suggested that assessments be performed to the extent possible remotely/virtually or delayed until such time that on-site visits can be resumed in order to continue participant monitoring in accordance with the protocol where possible. At each contact, participants will be interviewed to collect safety data. Key efficacy endpoint assessments should be performed if required and as feasible.

Modifications to protocol-required assessments may be permitted via COVID-19 Appendix after consultation with the participant, investigator, and the sponsor. Missed assessments/visits will be captured in the clinical trial management system for protocol deviations. Interruptions of test article wear or discontinuations of study interventions and withdrawal from the study should be documented with the prefix "COVID-19-related" in the case report form (CRF).

| Title: | Guidelines for CO | DVID-19 Risk Mitigation |
|-------------------------|-------------------|-------------------------|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

The sponsor will continue to monitor the conduct and progress of the clinical study, and any changes will be communicated to the sites and to the health authorities according to local guidance.

If a participant has tested positive for COVID-19, the investigator should contact the sponsor's responsible medical monitor to discuss initial plans for study intervention and follow-up. The medical monitor will notify the Safety Management Team of any subject(s) that have reported "COVID-19", "Asymptomatic COVID-19", or "Suspected COVID-19" adverse events within 24 hours of the notification.

Modifications made to the study conduct as a result of the COVID-19 pandemic will be summarized in the clinical study report.

COVID-19 screening procedures that may be mandated by local healthcare systems do not need to be reported as an amendment to the protocol even if done during clinical study visits.

#### 6.1 Monitoring Visits

When on-site monitoring by the sponsor is not feasible, the sponsor's site monitor will contact the study site to schedule remote visits. In such cases, on-site monitoring visits will resume when feasible, with increased frequency to address the source data verification backlog.

Even with staffing limitations during this COVID-19 pandemic, all routine operations related to clinical trials should be well-documented and archived as part of standard process. When conditions permit, all parties involved in this clinical trial should communicate relevant information in a timely manner so that all relevant parties remain sufficiently informed.

#### 6.1.1 Study Site Initiation:

During the period that this Work Instruction is in effect, Site Initiation Meetings and training of study site staff will be conducted remotely. The JJVCI study team will conduct training via Skype, Zoom, Microsoft Teams or similar software as well as utilize online training materials, as applicable. Study site training will be documented utilizing Site Initiation Report (Form Control No. ) per Study Site Initiation (Form Control No. ).

On-site visits may be considered when, for example, hands-on training or evaluation of site facilities is required. While on site, the Clinical Research Associate (CRA) will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

# 6.1.2 Interim Monitoring Visits (if applicable):

During the period that this Work Instruction is in effect, Interim Monitoring On-site visits will be kept to a minimum and include only those tasks that the CRA cannot perform remotely (e.g., source document verification, test article reconciliation, etc.).

To ensure data integrity during the conduct of all JJVC studies, clinical study teams will follow the study specific Clinical Monitoring Plan (Form Control No.

While on site, the CRA will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

| Title: | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | <b>Revision Number: 5</b> |

# 6.1.3 Study Site Closure:

During the period that this Work Instruction is in effect, the duration of the Study Site Closure Visit will be limited to tasks that the CRA cannot perform remotely (e.g., source document verification, test article final reconciliation and return, etc.).

| Title: | Guidelines for COVID-19 Risk M | itigation |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

## **Attachment A: Study Site Correspondence**

XXXX XX, 2020

# Re: COVID-19 Mitigation Plan, <<CR-xxxx/protocol title>>

Dear << Principal Investigator>> and Study Team,

Coronavirus (COVID-19) has impacted several communities and business activities over the past several months. While we work toward the successful conduct of clinical studies, our commitment continues to be the safety of patients, healthcare professionals, and to our communities.

Therefore, we would like to share the following revisions/additions related to the above referenced Johnson & Johnson Vision Care company sponsored clinical trial(s) you are currently working on or considering participation within.

## **Protocol:**

• Guidelines for COVID-19 Risk Mitigation provided in the Appendix section.

#### **Protocol Signature Page:**

 Will include a statement indicating the Principal Investigator agrees to conduct the study in compliance with all local, state, and governmental guidelines for COVID-19 risk mitigation.

# **Informed Consent:**

• Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed consent document.

# **COVID-19 Risk Control Checklist for Clinical Studies:**

• Will include COVID-19 risk control measures that are required to ensure the safety and health of subjects, site staff and monitors during the pandemic.

We want to encourage the need for open lines of communication about potential challenges you may foresee as the result of the current COVID-19 situation. Therefore, we encourage you to regularly connect with your respective Johnson & Johnson clinical study team (Clinical Research Associate (CRA), Lead CRA or Study Managers).

Thank you for your continued engagement, collaboration, and dedication to your study subjects during this challenging time.

Please file this letter in your site file study correspondence.

| Title: | Guidelines for COVID-19 Risk M | itigation |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

# **COVID-19 Risk Control Checklist (Attachment-B):**

Study Number Site Number Principal Investigator (PI) Name

The following COVID-19 risk control methods are required to conduct Johnson & Johnson Vison Care clinical studies. Please review the following requirements and Initial each requirement.

| PI Initials | General Site Safety Planning Measures |
|---|---|
| | Signage within site describing Risk Control methods |
| | Social Distancing practices throughout site (waiting rooms, lobby, exam rooms, etc.) |
| | Non-contact thermometer available to assess temperatures of staff and patients |
| | Training on patient flow and physical distancing in waiting room |
| | Establish longer time frame between patient appointments to reduce persons in the site |
| | Staff should receive job-specific training on PPE and demonstrate competency with selection and proper use of PPE and wear at all times during interactions with subjects (e.g., putting on and removing without self-contamination) |

| PI Initials | Site Staff Daily Safety Measures |
|---|---|
| | As part of routine practice, site staff should regularly monitor themselves for fever and symptoms |
| | of COVID-19, including temperature checks |
| | Any staff member (including non-study clinic staff and Investigators) showing signs of being sick |
| | or testing positive for COVID-19 must not be permitted to work on activity that may expose study |
| | related staff and subject and the Sponsor shall be informed |
| | NOTE: Inform JJVC in 24 hours of any COVID-19 cases and all potential exposure during |
| | the clinical study. |
| | Ensure that all staff wear a mask |
| | Gloves should be required when working directly with patients and changed between each patient |
| | Have staff thoroughly wash hands for at least 20 seconds or use an alcohol-based hand sanitizer |
| | when they arrive, before and after each patient, before eating and after using the bathroom. |
| | Cleaning and disinfection procedures for exam rooms and instruments or equipment between |
| | patients with gloves. |
| | Cleaning and disinfection procedures for commonly touched surfaces (doors, chairs, computers, |
| | phones, etc.) with gloves. |

| PI Initials | Before a Patient or Study Visit: |
|---|---|
| | Patients should be asked prior to entering the site about fever and respiratory illness and whether they or a family member have had contact with another person with confirmed COVID-19 in the past 14 days. Patients exhibiting signs of being sick should be rescheduled when their symptoms resolve. |
| | Instruct patients that companions should remain outside of the facility and not accompany the patient into the facility unless they are a parent/guardian of the patient or if they are a true caregiver and need to assist the patient |
| | Request the patient to call or text the office upon arrival so entrance to and movement through facility can be coordinated by site staff |

| Title: | Guidelines for CO | VID-19 Risk Mitigation |
|-------------------------|-------------------|------------------------|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | Revision Number: 5 |

| PI Initials | Patients Entering the site: |
|---|---|
| | Temperature checks utilizing a non-contact thermometer for all patients and companions entering |
| | the site. |
| | All patients and companions must wear cloth or disposable mask at all times in the site |
| | Maintain social distancing. Waiting rooms or lobbies should be as empty as possible. Advise |
| | seated patients to remain at least 6 feet from one another. |
| | Communal objects in (e.g. toys, reading materials, etc.) should be removed or cleaned regularly. |

I certify that I have read and agree to implement all the listed COVID-19 Risk Control Measures required for the conduct of Johnson & Johnson Vision Care studies.

Principal Investigator Signature and Date

| Title: | Guidelines for CO | Guidelines for COVID-19 Risk Mitigation | |
|---|---|---|---|
| <b>Document Type:</b> | | | |
| Document Number: | | | Revision Number: 5 |

# **RESOURCE LINKS**

# **US Resource Links**

OSHA Training

https://www.osha.gov/SLTC/covid-19/controlprevention.html

Personal Protective Equipment (PPE) Training

CDC: https://www.cdc.gov/coronavirus/2019-ncov/hcp/using-ppe.html

I&R Training

ACUVUE® LensAssist: https://www.acuvue.com/lensassist

• Clinic Preparedness Guides

CDC: <a href="https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinic-preparedness.html">https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinic-preparedness.html</a>
AOA: <a href="https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4="https://www.aoa.org/optometry-practice-reactivation-preparedness-guide">https://www.aoa.org/optometry-practice-reactivation-preparedness-guide</a>

• In-Office Disinfection of Multi-Patient Use Diagnostic Contact Lenses

<a href="https://www.gpli.info/wp-content/uploads/2020/03/2020-01-15-in-office-disinfecting-of-diagnostic-lenses.pdf">https://www.gpli.info/wp-content/uploads/2020/03/2020-01-15-in-office-disinfecting-of-diagnostic-lenses.pdf</a>

#### **OUS Resource Links**

- Updates on local regulations in Hong Kong https://www.coronavirus.gov.hk/eng/index.html
- Resumption of optical services in England: Letter from Matt Neligan and Poonam Sharma <a href="https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0601-reopening-of-optical-services-letter-17-june-2020.pdf">https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0601-reopening-of-optical-services-letter-17-june-2020.pdf</a>
- NHS Optical Letter
   <a href="https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0127-optical-letter-1-april-2020.pdf">https://www.england.nhs.uk/coronavirus/wp-content/uploads/sites/52/2020/04/C0127-optical-letter-1-april-2020.pdf</a>
- The College of Optometrists primary eye care COVID-19 guidance: Red phase <a href="https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-covid-19-guidance-for-optometrists.html">https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-covid-19-guidance-for-optometrists.html</a>
- The College of Optometrists COVID-19: College updates <a href="https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-2019-advice-for-optometrists.html#CollegeGuidelines">https://www.college-optometrists.org/the-college/media-hub/news-listing/coronavirus-2019-advice-for-optometrists.html#CollegeGuidelines</a>
- Infection Control Guidelines. (n.d.). Retrieved from Canadian Association Of Optometrists: https://opto.ca/sites/default/files/resources/documents/infection\_control\_guidelines\_2016.pdf
- Infection prevention and control for COVID-19: Interim guidance for outpatient and ambulatory care settings. (2020, May 23 May). Retrieved from Government of Canada: https://www.canada.ca/en/public-health/services/diseases/2019-novel-coronavirus-infection/guidance-documents/interim-guidance-outpatient-ambulatory-care-settings.html


| Title: | <b>Guidelines for COVID-19 Risk Mitigation</b> | |
|---|---|---|
| <b>Document Type:</b> | | |
| <b>Document Number:</b> | | <b>Revision Number: 5</b> |

- Information for Members On Coronavirus (COVID-19). (n.d.). Retrieved from Canadian Association Of Optometrists:
  - $https://opto.ca/sites/default/files/resources/documents/information\_for\_members\_on\_coronavirus.pdf$
- Coronavirus (COVID-19) resources for health professionals, including aged care providers, pathology providers and health care managers. (2020, September 24). Retrieved from Australian Government Department of Health:
  - https://www.health.gov.au/resources/collections/coronavirus-covid-19-resources-for-health-professionals-including-aged-care-providers-pathology-providers-and-health-care-managers
- Environmental Cleaning and Disinfection Principles for COVID-19. (n.d.). Retrieved from Australian Government Department of Health: https://www.health.gov.au/sites/default/files/documents/2020/03/environmental-cleaning-and-disinfection-principles-for-covid-19.pdf
- Infection control guidelines and advice. (n.d.). Retrieved from Optometry Australia: https://www.optometry.org.au/practice-professional-support/coronavirus-covid-19-what-optometrists-need-to-know/covid-19-clinical-advice/infection-control-guidelines-and-advice/


# Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

# PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6479 Protocol Title: Comparison of a Silicone Hydrogel Daily Disposable Multifocal Contact Lens to a Marketed Product

Version and Date: 3.0 15 March 2022

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155:2020,1 GCP and ICH guidelines,2 the Declaration of Helsinki,3 United States (US) Code of Federal Regulations (CFR),4 and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH2 regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH2 regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix J of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

| Principal<br>Investigator: | | |
|----------------------------|------------------------------------------|------|
| | Signature | Date |
| Institution/Site: | Name and Professional Position (Printed) | |
| | Institution/Site Name | |
| | Institution/Site Address | |